CLINICAL TRIAL: NCT03843359
Title: A Phase I First Time in Human Open Label Study of GSK3745417 Administered With and Without Anticancer Agents in Participants With Advanced Solid Tumors
Brief Title: A First Time in Human (FTIH) Study of GSK3745417 Administered to Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 208850
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Neoplasms
Keywords: GSK3745417; Dostarlimab; Anti-Programmed death receptor-1 (PD-1); Monoclonal antibody; Solid tumor; First time in human; Stimulator of Interferon Genes; STING
MeSH Terms: conditions — Neoplasms; Bites and Stings | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: In Part 1A, escalating doses of GSK3745417 will be evaluated and in Part 2A, escalating doses of GSK3745417 in combination with dostarlimab will be evaluated as guided by the Bayesian Logistic Regression Model (BLRM).
Masking Description: This will be an Open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1A: Participants receiving GSK3745417, Dose-escalation Cohort (Experimental)
  Interventions: Drug: GSK3745417
- Part 2A: Participants receiving GSK3745417 + dostarlimab, Dose escalation Cohort (Experimental)
  Interventions: Drug: GSK3745417; Drug: Dostarlimab

INTERVENTIONS:
Drug: GSK3745417 — GSK3745417 will be administered.
Drug: Dostarlimab — Dostarlimab will be administered.
  Arms: Part 2A: Participants receiving GSK3745417 + dostarlimab, Dose escalation Cohort

SUMMARY:
This study aims to evaluate the safety, tolerability, and preliminary clinical activity and establish a recommended dose of GSK3745417 administered alone (Part 1A) or co-administered (Part 2A) with dostarlimab in participants with refractory/relapsed solid tumors. Both parts will consist of a dose escalation phase.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be more than or equal to (>=)18 years of age.
* Participants with advanced/recurrent solid tumors, who have progressed on, be intolerant of, or ineligible for, all available therapies for which clinical benefit has been established.
* Histological or cytological documentation of an advanced solid tumor.
* Participants must provide a fresh biopsy.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
* Adequate organ function per protocol specifications.
* Male or female participants.
* Female participants are eligible to participate if they are not breastfeeding or pregnant (or intend to breastfeed or become pregnant). Women of childbearing potential must use a highly effective method of contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Active autoimmune disease that has required systemic disease modifying or immunosuppressive treatment within the last 2 years.
* Concurrent medical condition requiring the use of systemic immunosuppressive treatment within 28 days before the first dose of study treatment.
* Current unstable liver or biliary disease.
* History of vasculitis at any time prior to study treatment.
* Evidence or history of significant active bleeding or coagulation disorder.
* Active infection requiring systemic treatment, known human immunodeficiency virus infection, or positive test for hepatitis B surface antigen or hepatitis C.
* QT duration corrected for heart rate by Fridericia's formula (QTcF) more than (>)450 milliseconds (msec) or QTcF >480 msec for participants with bundle branch block.
* Recent history (within the past 6 months) of acute diverticulitis, inflammatory bowel disease, intra-abdominal abscess, or gastrointestinal obstruction.
* Recent history of allergen desensitization therapy within 4 weeks of starting study treatment.
* History or evidence of cardiovascular (CV) risk
* Recent (within the past 6 months) history of symptomatic pericarditis.
* History of idiopathic pulmonary fibrosis, interstitial lung disease, or organizing pneumonia, or evidence of active, non-infectious pneumonitis.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Recent history (within 6 months) of uncontrolled symptomatic ascites or pleural effusions.
* Prior treatment with the following agents:

  1. Stimulator of Interferon Genes (STING) agonist at any time.
  2. Anticancer therapy or investigational therapy or used an investigational device within 28 days or 5 half-lives of the drug, whichever is shorter.
  3. Checkpoint inhibitors, including Programmed death receptor-1 (PD-1), Programmed death Ligand-1 (PD-L1), PD-L2 and Cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) inhibitors within 28 days.
  4. Prior radiation therapy: permissible if at least 1 non-irradiated measurable lesion is available for assessment according to RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented.
* Pregnant and/or breast feeding participants or those who plan to become pregnant and/or breastfeed.
* Receipt of any live vaccine within 30 days of the start of study treatment.
* Prior allogeneic or autologous bone marrow transplantation or other solid organ transplantation.
* Major surgery less than or equal to (<=)28 days before the first dose of study treatment. Participants must have also fully recovered from any surgery (major or minor) and/or its complications before initiating study treatment.
* Participants with signs/symptoms suggestive of Coronavirus Disease-2019 (COVID-19) within 14 days of study entry, or with known exposure to COVID-19 within 14 days prior to study entry.
* Participants are excluded from Part 2A of the study if they have known hypersensitivity to dostarlimab or associated excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Houston, Texas, United States
- GSK Investigational Site, Melbourne, Victoria, Australia
- GSK Investigational Site, Toronto, Ontario, Canada
- France (2):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Tokyo, Japan
- GSK Investigational Site, Amsterdam, Netherlands
- GSK Investigational Site, Seoul, South Korea
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of 2 phases - Dose Escalation (Part 1A and Part 2A) and Dose Expansion (Part 1B and Part 2B). As pre-specified in protocol, dose expansion phases were not conducted following sponsor's decision to cease further enrolment into the study.
Pre-assignment Details: The results presented are based on the data cut-off date of 05 Apr 2024. Those participants still benefiting from study drug in the opinion of their treating physician continued to receive study drug in Post Analysis Continued Treatment (PACT) phase and their data will be reported after they stop receiving treatment as per protocol.
Groups:
- Part 1A: GSK3745417 0.1 mg (Q3W): Participants with advanced solid tumors received a 0.1 mg dose of GSK3745417 as an intravenous (IV) infusion every three weeks (Q3W) until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: GSK3745417 0.2 mg (Q3W): Participants with advanced solid tumors received a 0.2 mg dose of GSK3745417 as an IV infusion Q3W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: GSK3745417 0.1 mg (Q1W): Participants with Advanced Solid Tumors received 0.1 mg GSK3745417 as an IV infusion once a week (Q1W) until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: Japan GSK3745417 0.1 mg (Q1W): Japanese participants with Advanced Solid Tumors received 0.1 mg GSK3745417 as an IV infusion Q1W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: GSK3745417 0.2 mg (Q1W): Participants with Advanced Solid Tumors received 0.2 mg GSK3745417 as an IV infusion Q1W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: GSK3745417 0.4 mg (Q1W): Participants with Advanced Solid Tumors received 0.4 mg GSK3745417 as an IV infusion Q1W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis: Participants with Advanced Solid Tumors and effect of prophylaxis received 0.4 mg GSK3745417 as an IV infusion Q1W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.1 mg GSK3745417 as an IV infusion Q3W in combination with Dostarlimab 500 mg IV Q3W till Day 85 (Week 13), followed by 1000 mg IV every 6 weeks (Q6W) for subsequent doses until Day 722 or until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.2 mg GSK3745417 as an IV infusion Q3W in combination with Dostarlimab 500 mg IV Q3W till Day 85 (Week 13), followed by 1000 mg IV Q6W for subsequent doses until Day 722 or until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.1 mg GSK3745417 as an IV infusion Q1W in combination with Dostarlimab 500 mg IV Q3W till Day 85 (Week 13), followed by 1000 mg IV Q6W for subsequent doses until Day 722 or until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.1 mg GSK3745417 as an IV infusion Q1W in combination with Dostarlimab 500 mg IV Q3W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier. Additionally, for participants in this arm T-cell activation through Positron Emission Tomography (PET) imaging of 18F-labeled analog of arabinofuranosyl guanine ([18F]F-AraG) and the biodistribution of radiolabeled GSK3745417 were performed.
- Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.2 mg GSK3745417 as an IV infusion Q1W combination with Dostarlimab 500 mg IV Q3W till Day 85 (Week 13), followed by 1000 mg IV Q6W for subsequent doses until Day 722 or until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier.
- Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab: Participants with Advanced Solid Tumors received 0.2 mg GSK3745417 as an IV infusion Q1W in combination with Dostarlimab 500 mg IV Q3W until disease progression, death, the onset of unacceptable toxicity (including meeting liver chemistry stopping criteria), withdrawal of consent, or upto 2 years, whichever occurred earlier. Additionally, for participants in this arm T-cell activation through PET imaging of [18F]F-AraG and the biodistribution of radiolabeled GSK3745417 were performed.
- Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab: Participants with advanced solid tumors who received GSK3745417 monotherapy in Part 1A, upon disease progression, crossed over received 0.1 mg GSK3745417 as an IV infusion Q3W in combination with Dostarlimab 500 mg IV Q3W, followed by 1000 mg IV every 6 weeks (Q6W) until 30.3 weeks.
- Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab: Participants with advanced solid tumors who received GSK3745417 monotherapy in Part 1A, upon disease progression, crossed over and received 0.2 mg GSK3745417 as an IV infusion Q3W in combination with Dostarlimab 500 mg IV Q3W, followed by 1000 mg IV Q6W until 30.3 weeks.
- Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab: Participants with advanced solid tumors who received GSK3745417 monotherapy in Part 1A, upon disease progression, crossed over and received 0.1 mg GSK3745417 as an IV infusion Q1W in combination with Dostarlimab 500 mg IV Q3W followed by 1000 mg IV Q6W until 30.3 weeks.
Period: Escalation Phase
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W) | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Started | 3 | 6 | 14 | 2 | 19 | 10 | 9 | 4 | 12 | 4 | 3 | 10 | 1 | 0 | 0 | 0
All Treated Population (All participants who received at least one dose of GSK3745417) | 3 | 6 | 14 | 2 | 19 | 10 | 9 | 4 | 12 | 4 | 3 | 10 | 1 | 0 | 0 | 0
Dose-Limiting Toxicities (DLT)Evaluable Population (All Treated population who completed at least 21 or 29 days of DLT period or discontinued from treatment within 21 or 29 days due to an AE meeting the definition of a DLT) | 3 | 4 | 4 | 2 | 9 | 9 | 0 | 4 | 9 | 4 | 0 | 4 | 0 | 0 | 0 | 0
Pharmacokinetic (PK) Population (All participants from the All-Treated Population for whom a PK sample were obtained and analyzed.) | 3 | 6 | 14 | 2 | 19 | 10 | 9 | 4 | 12 | 4 | 3 | 10 | 1 | 0 | 0 | 0
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 3 (3 participants died) | 5 (5 participants died) | 6 (6 participants died) | 1 (1 participant completed follow-up) | 15 (1 participant completed follow-up and 14 participants died) | 9 (2 participants completed follow-up and 7 participants died) | 8 (8 participants died) | 4 (1 participants completed follow-up and 3 participants died) | 8 (8 participants died) | 4 (4 participants died) | 3 (1 participant completed follow-up and 2 participants died) | 9 (1 participant completed follow-up and 8 participants died) | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 8 | 1 | 4 | 1 | 1 | 0 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator site closed | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing at the time of analysis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Participants were crossed over OR were re-treated following progression | 0 | 0 | 7 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Crossover
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W) | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (As prespecified in protocol, participants enrolled in Part 1A (GSK3745417 monotherapy) upon disease progression were allowed to receive GSK3745417 in combination with dostarlimab (defined as crossover)) | 4 (As prespecified in protocol, participants enrolled in Part 1A (GSK3745417 monotherapy) upon disease progression were allowed to receive GSK3745417 in combination with dostarlimab (defined as crossover)) | 5 (As prespecified in protocol, participants enrolled in Part 1A (GSK3745417 monotherapy) upon disease progression were allowed to receive GSK3745417 in combination with dostarlimab (defined as crossover))
All Treated Population (All participants who received at least one dose of GSK3745417) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5
Pharmacokinetic (PK) Population (All participants from the All-Treated Population for whom a PK sample were obtained and analyzed.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (1 participant completed follow-up and 1 participant died) | 2 (2 participants died)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator site closed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Ongoing at the time of analysis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W) | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab | Total
Number analyzed (Participants) | 3 | 6 | 14 | 2 | 19 | 10 | 9 | 4 | 12 | 4 | 3 | 10 | 1 | 97
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 50.0 (1.73) | 46.8 (17.81) | 55.8 (11.44) | 66.0 (2.83) | 56.5 (15.13) | 53.3 (11.41) | 51.3 (9.08) | 66.3 (5.80) | 55.5 (12.21) | 54.5 (7.14) | 61.7 (12.50) | 58.0 (10.45) | NA (NA) — No data was reported to maintain participant (0<n<2) confidentiality and privacy. | 55.5 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 7 | 0 | 9 | 7 | 7 | 4 | 4 | 2 | 0 | 5 | 1 | 50
  Male | 2 | 3 | 7 | 2 | 10 | 3 | 2 | 0 | 8 | 2 | 3 | 5 | 0 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 14 | 2 | 19 | 10 | 9 | 4 | 12 | 4 | 3 | 10 | 1 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 6 | 13 | 0 | 19 | 10 | 9 | 3 | 10 | 3 | 0 | 8 | 0 | 84
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part 1A: Number of Participants Achieving Dose-limiting Toxicity (DLT) Following Administration of GSK3745417 Alone (Q1W)
Description: AE is DLT if deemed clinically relevant,attributed to study intervention & met DLT criteria:CytokineReleaseSyndrome (CRS) (Grade(G) 3/4);Liver Toxicity: ALT≥3xULN + bilirubin≥2xULN/INR>1.5, ALT≥5x ULN+≥2x baseline with liver,metastases/tumor infiltration or HCC;G≥3 non-hematologic exceptions: Transient lab abnormalities, CRS≤G2,Controlled diarrhea,Resolving nausea/vomiting,Alopecia,G3 fatigue<7 days,G3 headache resolving in 24 hrs;G≥3 immune-related toxicity unresolved in 8 days despite therapy and G≥3 infusion reactions included;Other toxicities: G≥2 uveitis, Unresolved eye pain/blurred vision in 2 wks,Endocrine toxicity needing hormone replacement,Colitis/diarrhea unresolved for ≥7Days despite steroids,ICANS;Hematologic toxicity includes: Neutropenia(G4 ≥7Days or G3/4 with infection/febrile neutropenia),Thrombocytopenia (G4/G3 with bleeding/transfusion),Anemia (G4/G3 needing transfusion);Other events deemed DLTs by the investigator and GSK Medical Monitor per NCI-CTCAE v5.0
Time Frame: Up to 21 Days
Population: DLT Evaluable population included All Treated population who completed at least 21 days of DLT period or discontinued from treatment within 21 days due to an AE meeting the definition of a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W)
Number analyzed (Participants) | 4 | 2 | 9 | 9
Participants | 0 | 0 | 0 | 2

2. Primary Outcome: Parts 1A: Number of Participants Achieving DLT Following Administration of GSK3745417 Alone (Q3W)
Description: as for outcome 1
Time Frame: Up to 29 Days
Population: DLT Evaluable population included All Treated population who completed at least 29 days of DLT period or discontinued from treatment within 29 days due to an AE meeting the definition of a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W)
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

3. Primary Outcome: Parts 2A: Number of Participants Achieving DLT Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 1
Time Frame: Up to 29 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

4. Primary Outcome: Parts 2A: Number of Participants Achieving Dose-limiting Toxicity (DLT) Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 1
Time Frame: Up to 29 Days
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 4 | 9
Participants | 0 | 0

5. Primary Outcome: Parts 1A: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (STEAEs) by Severity
Description: AE is any untoward medical occurrence in clinical investigation participant, temporally associated with the use of medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. AEs were graded by the investigator according to National Cancer Institute Common Terminology Criteria for AE (NCI-CTCAE) (version 5.0):G1=Mild,G2=Moderate,G3=Severe or medically significant but not immediately life-threatening,G4=Life-threatening consequences,G5=Death related AE.
Time Frame: Up to approximately 62 weeks
Population: All treated population included all participants who received at least one dose of GSK3745417. Each participant was counted only once, based on the highest grade they experienced across all adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W) | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis
Number analyzed (Participants) | 3 | 6 | 14 | 2 | 19 | 10 | 9
Participants
  TEAEs, Grade 1 | 2 | 0 | 2 | 1 | 5 | 0 | 1
  TEAEs, Grade 2 | 0 | 4 | 6 | 1 | 5 | 5 | 3
  TEAEs, Grade 3 | 0 | 1 | 6 | 0 | 8 | 5 | 5
  TEAEs, Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  TEAEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  STEAEs, Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  STEAEs, Grade 2 | 0 | 0 | 2 | 0 | 2 | 3 | 0
  STEAEs, Grade 3 | 0 | 0 | 2 | 0 | 5 | 0 | 2
  STEAEs, Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  STEAEs, Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Parts 2A: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (STEAEs) by Severity
Description: AE is any untoward medical occurrence in clinical investigation participant, temporally associated with the use of medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. SAEs are subset of AEs. TEAE is an event that emerges during treatment having been absent pretreatment or worsens relative to the pretreatment state. AEs were graded by the investigator according to NCI-CTCAE v5.0: G1=Mild, G2=Moderate, G3=Severe or medically significant but not immediately life-threatening, G4=Life-threatening consequences, G5=Death related AE.
Time Frame: Up to approximately 93 weeks
Population: All treated population. Each participant was counted only once, based on the highest grade they experienced across all adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 12 | 4 | 3 | 10 | 1
Participants
  TEAEs, Grade 1 | 1 | 3 | 0 | 1 | 1 | 0
  TEAEs, Grade 2 | 2 | 2 | 0 | 0 | 5 | 1
  TEAEs, Grade 3 | 1 | 4 | 4 | 2 | 2 | 0
  TEAEs, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0
  TEAEs, Grade 5 | 0 | 2 | 0 | 0 | 2 | 0
  STEAEs, Grade 1 | 0 | 0 | 0 | 0 | 0 | 1
  STEAEs, Grade 2 | 0 | 1 | 0 | 1 | 0 | 0
  STEAEs, Grade 3 | 1 | 2 | 3 | 1 | 2 | 0
  STEAEs, Grade 4 | 0 | 1 | 0 | 0 | 0 | 0
  STEAEs, Grade 5 | 0 | 2 | 0 | 0 | 2 | 0

7. Primary Outcome: Crossover Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Treatment-emergent Adverse Events (STEAEs) by Severity
Description: as for outcome 6
Time Frame: Up to 30.3 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 1 | 4 | 5
Participants
  TEAEs, Grade 1 | 0 | 1 | 1
  TEAEs, Grade 2 | 1 | 0 | 3
  TEAEs, Grade 3 | 0 | 2 | 1
  TEAEs, Grade 4 | 0 | 0 | 0
  TEAEs, Grade 5 | 0 | 0 | 0
  STEAEs, Grade 1 | 0 | 0 | 0
  STEAEs, Grade 2 | 0 | 0 | 0
  STEAEs, Grade 3 | 0 | 1 | 1
  STEAEs, Grade 4 | 0 | 0 | 0
  STEAEs, Grade 5 | 0 | 0 | 0

8. Secondary Outcome: Part 1A: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 Alone (Q1W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Pre-dose on weeks(W) 1-6,9,10,12,19,55;end of infusion(EOI)+5minute(min) on W 1-6, 9,10,12,19,55;EOI+4 hour(HR)/8 HR on W 1-6, 9, 10, 12, 19;EOI+15min/30min/45min/1HR on W 1-6, 9,12;EOI+24HR on W 1-6, 9,10,12; EOI+2HR on W 1-6,9,10,12,19,55
Population: Pharmacokinetic (PK) population included all participants from the All Treated Population for whom at least one PK sample was obtained and analyzed. The number analyzed for each timepoint reflects the number of participants from the Overall PK population with a non-missing value at the specified time point.
Measure: Median (Full Range); unit: Nanogram/ millilitre (ng/mL)
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis
Number analyzed (Participants) | 14 | 2 | 19 | 10 | 9
Nanogram/ millilitre (ng/mL)
  WEEK1, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK1, EOI+5MIN | 21.365 [9.750 to 49.540] | 15.000 [0.000 to 30.000] | 44.700 [25.800 to 90.770] | 103.550 [75.450 to 145.080] | 111.655 [79.945 to 132.755]
  WEEK1, EOI+15MIN | 18.880 [8.830 to 40.940] | 18.590 [8.580 to 28.600] | 40.700 [25.600 to 95.960] | 90.640 [64.340 to 119.480] | 96.102 [53.635 to 147.868]
  WEEK1, EOI+30MIN | 15.800 [7.540 to 40.680] | 17.050 [8.700 to 25.400] | 36.000 [22.300 to 91.110] | 83.075 [43.280 to 102.680] | 78.439 [32.800 to 123.949]
  WEEK1, EOI+45MIN | 13.150 [5.890 to 33.470] | 14.365 [4.830 to 23.900] | 31.420 [15.300 to 78.940] | 70.485 [39.880 to 89.590] | 66.000 [23.487 to 110.269]
  WEEK1, EOI+1HR: number analyzed (Participants) | 14 | 1 | 19 | 10 | 9
  WEEK1, EOI+1HR | 10.580 [5.030 to 33.620] | 21.300 [21.300 to 21.300] | 29.000 [11.200 to 75.950] | 62.310 [28.870 to 92.810] | 59.051 [17.933 to 124.574]
  WEEK1, EOI+2HR | 6.090 [2.440 to 18.210] | 34.100 [16.400 to 51.800] | 16.200 [6.370 to 44.710] | 32.970 [6.420 to 74.810] | 39.142 [3.596 to 105.515]
  WEEK1, EOI+4HR | 2.030 [0.000 to 12.490] | 24.690 [8.580 to 40.800] | 6.000 [0.000 to 27.300] | 11.380 [0.000 to 65.420] | 12.886 [0.701 to 67.719]
  WEEK1, EOI+8HR | 0.195 [0.000 to 4.620] | 17.930 [4.560 to 31.300] | 0.338 [0.000 to 19.600] | 0.000 [0.000 to 37.960] | 2.200 [0.286 to 49.586]
  WEEK1, EOI+24HR: number analyzed (Participants) | 14 | 2 | 19 | 9 | 9
  WEEK1, EOI+24HR | 0.000 [0.000 to 0.488] | 3.460 [0.939 to 5.980] | 0.000 [0.000 to 6.790] | 0.000 [0.000 to 0.000] | 0.700 [0.000 to 6.781]
  WEEK2, PREDOSE: number analyzed (Participants) | 12 | 2 | 18 | 8 | 9
  WEEK2, PREDOSE | 0.000 [0.000 to 0.020] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 1.690] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.209]
  WEEK2, EOI+5MIN: number analyzed (Participants) | 14 | 2 | 18 | 9 | 9
  WEEK2, EOI+5MIN | 23.550 [14.600 to 42.090] | 21.350 [13.300 to 29.400] | 49.810 [7.710 to 80.800] | 119.990 [69.420 to 162.650] | 111.450 [71.438 to 153.211]
  WEEK2, EOI+15MIN: number analyzed (Participants) | 4 | 0 | 9 | 9 | 9
  WEEK2, EOI+15MIN | 21.110 [19.340 to 38.180] |  | 45.700 [30.210 to 73.210] | 99.730 [58.350 to 137.590] | 94.602 [67.624 to 136.044]
  WEEK2, EOI+30MIN: number analyzed (Participants) | 4 | 0 | 9 | 9 | 9
  WEEK2, EOI+30MIN | 16.790 [16.560 to 37.000] |  | 36.370 [23.510 to 69.480] | 92.780 [47.530 to 135.670] | 80.173 [38.867 to 130.765]
  WEEK2, EOI+45MIN: number analyzed (Participants) | 4 | 0 | 9 | 9 | 9
  WEEK2, EOI+45MIN | 15.735 [13.110 to 32.440] |  | 31.750 [21.090 to 67.680] | 79.810 [37.510 to 136.940] | 75.977 [31.154 to 114.318]
  WEEK2, EOI+1HR: number analyzed (Participants) | 4 | 0 | 9 | 9 | 9
  WEEK2, EOI+1HR | 14.545 [10.540 to 30.160] |  | 31.230 [19.790 to 63.710] | 73.750 [23.800 to 135.510] | 74.026 [22.289 to 111.132]
  WEEK2, EOI+2HR: number analyzed (Participants) | 14 | 2 | 18 | 9 | 9
  WEEK2, EOI+2HR | 7.880 [4.620 to 23.280] | 13.400 [13.300 to 13.500] | 15.695 [4.390 to 45.830] | 45.560 [12.840 to 104.090] | 50.148 [5.842 to 97.944]
  WEEK2, EOI+4HR: number analyzed (Participants) | 14 | 2 | 18 | 9 | 9
  WEEK2, EOI+4HR | 2.490 [0.000 to 14.260] | 7.320 [6.730 to 7.910] | 8.150 [0.000 to 31.700] | 17.490 [0.000 to 86.110] | 20.212 [1.238 to 79.302]
  WEEK2, EOI+8HR: number analyzed (Participants) | 14 | 2 | 18 | 9 | 9
  WEEK2, EOI+8HR | 0.381 [0.000 to 5.670] | 2.840 [2.660 to 3.020] | 0.438 [0.000 to 23.900] | 0.000 [0.000 to 60.670] | 7.987 [0.393 to 38.692]
  WEEK2, EOI+24HR: number analyzed (Participants) | 14 | 2 | 18 | 9 | 9
  WEEK2, EOI+24HR | 0.067 [0.000 to 4.580] | 0.516 [0.465 to 0.566] | 0.000 [0.000 to 11.400] | 0.000 [0.000 to 21.740] | 1.129 [0.000 to 7.613]
  WEEK3, PREDOSE: number analyzed (Participants) | 14 | 2 | 17 | 8 | 4
  WEEK3, PREDOSE | 0.000 [0.000 to 2.080] | 0.665 [0.000 to 1.330] | 0.000 [0.000 to 2.240] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.135]
  WEEK3, EOI+5MIN: number analyzed (Participants) | 14 | 2 | 17 | 8 | 6
  WEEK3, EOI+5MIN | 24.245 [0.000 to 43.900] | 9.390 [2.280 to 16.500] | 49.010 [24.000 to 94.440] | 101.655 [64.490 to 131.300] | 121.546 [70.878 to 139.062]
  WEEK3, EOI+15MIN: number analyzed (Participants) | 4 | 0 | 9 | 8 | 6
  WEEK3, EOI+15MIN | 27.620 [0.000 to 42.040] |  | 44.120 [36.050 to 75.680] | 97.570 [58.290 to 120.930] | 104.424 [57.080 to 117.498]
  WEEK3, EOI+30MIN: number analyzed (Participants) | 4 | 0 | 9 | 8 | 6
  WEEK3, EOI+30MIN | 25.495 [0.000 to 36.620] |  | 36.790 [29.720 to 60.530] | 90.085 [48.580 to 114.000] | 85.103 [44.011 to 118.110]
  WEEK3, EOI+45MIN: number analyzed (Participants) | 4 | 0 | 9 | 8 | 6
  WEEK3, EOI+45MIN | 23.095 [0.000 to 37.000] |  | 34.510 [24.970 to 55.420] | 76.765 [42.740 to 110.030] | 69.923 [29.713 to 100.740]
  WEEK3, EOI+1HR: number analyzed (Participants) | 4 | 0 | 9 | 8 | 6
  WEEK3, EOI+1HR | 21.055 [0.000 to 30.990] |  | 32.030 [21.590 to 61.020] | 63.890 [28.690 to 101.890] | 56.589 [21.538 to 93.551]
  WEEK3, EOI+2HR: number analyzed (Participants) | 14 | 2 | 17 | 8 | 6
  WEEK3, EOI+2HR | 10.020 [0.000 to 24.840] | 8.460 [0.319 to 16.600] | 17.600 [5.520 to 38.780] | 41.550 [14.870 to 72.560] | 32.906 [6.756 to 66.786]
  WEEK3, EOI+4HR: number analyzed (Participants) | 14 | 2 | 17 | 8 | 6
  WEEK3, EOI+4HR | 2.970 [0.000 to 13.980] | 5.072 [0.244 to 9.900] | 8.480 [0.000 to 33.800] | 14.945 [0.000 to 57.790] | 14.279 [1.563 to 32.725]
  WEEK3, EOI+8HR: number analyzed (Participants) | 14 | 1 | 16 | 8 | 6
  WEEK3, EOI+8HR | 0.462 [0.000 to 8.930] | 5.480 [5.480 to 5.480] | 0.236 [0.000 to 20.500] | 2.845 [0.000 to 32.450] | 1.944 [0.344 to 8.853]
  WEEK3, EOI+24HR: number analyzed (Participants) | 14 | 1 | 17 | 8 | 6
  WEEK3, EOI+24HR | 0.054 [0.000 to 2.240] | 1.020 [1.020 to 1.020] | 0.000 [0.000 to 10.000] | 0.000 [0.000 to 11.610] | 0.459 [0.111 to 2.797]
  WEEK4, PREDOSE: number analyzed (Participants) | 12 | 2 | 17 | 9 | 7
  WEEK4, PREDOSE | 0.000 [0.000 to 0.508] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 2.990] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK4, EOI+5MIN: number analyzed (Participants) | 13 | 2 | 17 | 9 | 7
  WEEK4, EOI+5MIN | 22.730 [3.240 to 40.280] | 27.850 [23.100 to 32.600] | 49.095 [9.840 to 99.630] | 106.260 [77.200 to 157.530] | 112.175 [80.304 to 156.837]
  WEEK4, EOI+15MIN: number analyzed (Participants) | 13 | 0 | 15 | 9 | 7
  WEEK4, EOI+15MIN | 20.300 [4.950 to 35.770] |  | 41.540 [12.420 to 75.620] | 99.440 [57.180 to 131.180] | 102.480 [64.598 to 139.072]
  WEEK4, EOI+30MIN: number analyzed (Participants) | 13 | 0 | 15 | 9 | 7
  WEEK4, EOI+30MIN | 16.800 [3.870 to 33.540] |  | 33.500 [11.100 to 68.820] | 92.590 [49.600 to 123.280] | 90.573 [42.598 to 123.215]
  WEEK4, EOI+45MIN: number analyzed (Participants) | 13 | 0 | 15 | 9 | 7
  WEEK4, EOI+45MIN | 13.380 [3.330 to 28.270] |  | 31.300 [9.500 to 61.460] | 85.550 [38.820 to 120.770] | 68.947 [34.245 to 112.398]
  WEEK4, EOI+1HR: number analyzed (Participants) | 13 | 0 | 15 | 9 | 7
  WEEK4, EOI+1HR | 11.400 [1.020 to 27.590] |  | 28.030 [13.900 to 54.720] | 66.970 [28.640 to 115.460] | 64.737 [23.292 to 119.650]
  WEEK4, EOI+2HR: number analyzed (Participants) | 13 | 2 | 17 | 9 | 7
  WEEK4, EOI+2HR | 6.990 [0.000 to 19.260] | 14.000 [11.700 to 16.300] | 17.320 [5.790 to 52.020] | 31.510 [10.400 to 107.260] | 38.423 [5.331 to 68.771]
  WEEK4, EOI+4HR: number analyzed (Participants) | 13 | 2 | 17 | 9 | 7
  WEEK4, EOI+4HR | 1.850 [0.000 to 14.240] | 8.605 [6.710 to 10.500] | 7.620 [0.000 to 34.600] | 10.710 [0.000 to 95.570] | 13.288 [1.373 to 37.803]
  WEEK4, EOI+8HR: number analyzed (Participants) | 13 | 1 | 16 | 9 | 7
  WEEK4, EOI+8HR | 0.391 [0.000 to 5.270] | 4.020 [4.020 to 4.020] | 0.129 [0.000 to 25.900] | 8.370 [0.000 to 57.020] | 2.564 [0.362 to 9.556]
  WEEK4, EOI+24HR: number analyzed (Participants) | 13 | 1 | 15 | 9 | 7
  WEEK4, EOI+24HR | 0.000 [0.000 to 1.070] | 0.791 [0.791 to 0.791] | 0.000 [0.000 to 12.700] | 0.000 [0.000 to 19.210] | 0.686 [0.114 to 3.722]
  WEEK5, PREDOSE: number analyzed (Participants) | 11 | 2 | 14 | 7 | 7
  WEEK5, PREDOSE | 0.000 [0.000 to 0.195] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 2.970] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.137]
  WEEK5, EOI+5MIN: number analyzed (Participants) | 11 | 2 | 14 | 7 | 7
  WEEK5, EOI+5MIN | 19.480 [7.720 to 27.600] | 21.350 [16.000 to 26.700] | 47.173 [26.800 to 87.170] | 113.140 [66.480 to 162.700] | 112.617 [85.635 to 137.264]
  WEEK5, EOI+15MIN: number analyzed (Participants) | 3 | 0 | 8 | 7 | 7
  WEEK5, EOI+15MIN | 17.260 [15.400 to 18.550] |  | 42.492 [38.480 to 78.400] | 106.120 [57.190 to 150.860] | 94.482 [72.447 to 129.269]
  WEEK5, EOI+30MIN: number analyzed (Participants) | 3 | 0 | 8 | 7 | 7
  WEEK5, EOI+30MIN | 15.290 [12.650 to 19.120] |  | 33.345 [29.640 to 73.610] | 85.740 [43.400 to 137.520] | 76.850 [51.081 to 112.129]
  WEEK5, EOI+45MIN: number analyzed (Participants) | 3 | 0 | 8 | 7 | 7
  WEEK5, EOI+45MIN | 14.090 [10.100 to 15.940] |  | 27.900 [23.750 to 72.770] | 92.490 [36.760 to 106.330] | 70.156 [46.092 to 105.535]
  WEEK5, EOI+1HR: number analyzed (Participants) | 3 | 0 | 8 | 7 | 7
  WEEK5, EOI+1HR | 12.510 [8.940 to 14.180] |  | 25.885 [22.437 to 60.580] | 69.760 [34.670 to 102.530] | 69.849 [29.221 to 100.886]
  WEEK5, EOI+2HR: number analyzed (Participants) | 11 | 2 | 13 | 7 | 7
  WEEK5, EOI+2HR | 7.370 [0.000 to 12.500] | 14.000 [11.300 to 16.700] | 14.350 [6.290 to 41.800] | 47.890 [15.200 to 84.870] | 49.617 [9.674 to 78.627]
  WEEK5, EOI+4HR: number analyzed (Participants) | 11 | 2 | 14 | 7 | 7
  WEEK5, EOI+4HR | 1.620 [0.000 to 7.760] | 8.010 [6.200 to 9.820] | 5.495 [0.000 to 34.500] | 23.080 [0.000 to 51.940] | 22.082 [2.296 to 52.873]
  WEEK5, EOI+8HR: number analyzed (Participants) | 11 | 1 | 14 | 7 | 7
  WEEK5, EOI+8HR | 0.397 [0.000 to 4.200] | 3.470 [3.470 to 3.470] | 0.746 [0.000 to 25.900] | 6.120 [0.000 to 39.080] | 2.599 [0.492 to 21.474]
  WEEK5, EOI+24HR: number analyzed (Participants) | 11 | 1 | 14 | 7 | 7
  WEEK5, EOI+24HR | 0.000 [0.000 to 0.920] | 0.856 [0.856 to 0.856] | 0.000 [0.000 to 12.200] | 0.000 [0.000 to 16.490] | 0.752 [0.137 to 6.687]
  WEEK6, PREDOSE: number analyzed (Participants) | 11 | 2 | 10 | 5 | 4
  WEEK6, PREDOSE | 0.000 [0.000 to 0.133] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 3.410] | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK6, EOI+5MIN: number analyzed (Participants) | 12 | 2 | 9 | 5 | 4
  WEEK6, EOI+5MIN | 18.575 [8.130 to 26.600] | 18.650 [18.600 to 18.700] | 58.328 [17.800 to 90.060] | 106.730 [65.440 to 153.340] | 102.851 [99.360 to 127.991]
  WEEK6, EOI+15MIN: number analyzed (Participants) | 10 | 0 | 8 | 5 | 4
  WEEK6, EOI+15MIN | 16.120 [6.870 to 25.200] |  | 37.845 [15.400 to 78.220] | 121.300 [57.500 to 124.410] | 86.413 [79.637 to 110.036]
  WEEK6, EOI+30MIN: number analyzed (Participants) | 10 | 0 | 8 | 5 | 4
  WEEK6, EOI+30MIN | 14.750 [5.760 to 21.700] |  | 32.860 [13.700 to 75.200] | 78.930 [45.740 to 107.870] | 62.879 [58.925 to 90.275]
  WEEK6, EOI+45MIN: number analyzed (Participants) | 10 | 0 | 8 | 5 | 4
  WEEK6, EOI+45MIN | 12.550 [4.890 to 20.000] |  | 28.320 [13.100 to 77.710] | 87.250 [37.250 to 97.940] | 47.588 [38.173 to 90.417]
  WEEK6, EOI+1HR: number analyzed (Participants) | 10 | 0 | 8 | 5 | 4
  WEEK6, EOI+1HR | 11.950 [0.000 to 17.400] |  | 30.325 [11.400 to 65.470] | 76.440 [35.500 to 82.840] | 40.026 [35.272 to 75.498]
  WEEK6, EOI+2HR: number analyzed (Participants) | 12 | 2 | 10 | 5 | 4
  WEEK6, EOI+2HR | 5.930 [0.000 to 11.960] | 11.500 [11.300 to 11.700] | 17.485 [5.700 to 61.870] | 41.620 [18.180 to 58.650] | 15.285 [13.620 to 53.502]
  WEEK6, EOI+4HR: number analyzed (Participants) | 12 | 2 | 10 | 5 | 4
  WEEK6, EOI+4HR | 2.085 [0.000 to 8.480] | 6.190 [6.160 to 6.220] | 7.630 [0.000 to 42.100] | 13.200 [0.000 to 38.270] | 3.917 [3.691 to 36.777]
  WEEK6, EOI+8HR: number analyzed (Participants) | 12 | 0 | 10 | 5 | 4
  WEEK6, EOI+8HR | 0.473 [0.000 to 5.710] |  | 1.642 [0.000 to 35.000] | 0.000 [0.000 to 23.100] | 0.935 [0.732 to 12.042]
  WEEK6, EOI+24HR: number analyzed (Participants) | 11 | 0 | 10 | 5 | 4
  WEEK6, EOI+24HR | 0.000 [0.000 to 0.711] |  | 0.201 [0.000 to 17.800] | 0.000 [0.000 to 8.670] | 0.269 [0.203 to 1.786]
  WEEK9, PREDOSE: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, PREDOSE | 0.000 [0.000 to 12.690] |  | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 22.160] | 0.145 [0.000 to 0.206]
  WEEK9, EOI+5MIN: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+5MIN | 22.990 [11.770 to 26.810] |  | 43.295 [27.250 to 59.340] | 126.020 [74.630 to 173.550] | 98.752 [84.687 to 107.093]
  WEEK9, EOI+15MIN: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+15MIN | 17.340 [10.410 to 22.360] |  | 46.830 [43.320 to 50.340] | 116.030 [63.120 to 129.190] | 90.104 [65.049 to 118.578]
  WEEK9, EOI+30MIN: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+30MIN | 11.570 [9.050 to 20.500] |  | 38.160 [36.160 to 40.160] | 108.240 [56.100 to 115.620] | 83.767 [47.615 to 94.767]
  WEEK9, EOI+45MIN: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+45MIN | 8.730 [7.440 to 15.990] |  | 30.000 [23.950 to 36.050] | 85.520 [47.830 to 101.440] | 80.187 [37.837 to 87.354]
  WEEK9, EOI+1HR: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+1HR | 7.700 [6.760 to 12.680] |  | 25.965 [24.910 to 27.020] | 75.860 [36.360 to 100.500] | 70.788 [25.646 to 85.403]
  WEEK9, EOI+2HR: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+2HR | 0.000 [0.000 to 7.240] |  | 14.675 [13.170 to 16.180] | 36.110 [15.410 to 50.650] | 48.390 [9.266 to 54.623]
  WEEK9, EOI+4HR: number analyzed (Participants) | 3 | 0 | 2 | 3 | 3
  WEEK9, EOI+4HR | 0.000 [0.000 to 0.000] |  | 3.020 [0.000 to 6.040] | 20.740 [6.060 to 27.760] | 37.657 [3.645 to 41.961]
  WEEK9, EOI+8HR: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK9, EOI+8HR | 0.000 [0.000 to 0.000] |  |  |  |
  WEEK9, EOI+24HR: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK9, EOI+24HR | 0.000 [0.000 to 0.000] |  |  |  |
  WEEK10, PREDOSE: number analyzed (Participants) | 6 | 1 | 2 | 0 | 0
  WEEK10, PREDOSE | 0.000 [0.000 to 3.840] | 0.000 [0.000 to 0.000] | 3.150 [0.000 to 6.300] |  |
  WEEK10, EOI+5MIN: number analyzed (Participants) | 6 | 1 | 2 | 0 | 0
  WEEK10, EOI+5MIN | 17.250 [8.120 to 34.600] | 27.400 [27.400 to 27.400] | 71.450 [70.800 to 72.100] |  |
  WEEK10, EOI+2HR: number analyzed (Participants) | 6 | 1 | 2 | 0 | 0
  WEEK10, EOI+2HR | 6.210 [4.280 to 10.100] | 12.700 [12.700 to 12.700] | 38.650 [24.400 to 52.900] |  |
  WEEK10, EOI+4HR: number analyzed (Participants) | 6 | 1 | 2 | 0 | 0
  WEEK10, EOI+4HR | 2.205 [1.140 to 7.000] | 7.400 [7.400 to 7.400] | 25.150 [7.800 to 42.500] |  |
  WEEK10, EOI+8HR: number analyzed (Participants) | 5 | 0 | 1 | 0 | 0
  WEEK10, EOI+8HR | 0.462 [0.255 to 1.570] |  | 2.300 [2.300 to 2.300] |  |
  WEEK10, EOI+24HR: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK10, EOI+24HR | 0.268 [0.268 to 0.268] |  |  |  |
  WEEK12, PREDOSE: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, PREDOSE | 0.000 [0.000 to 0.000] |  | 0.000 [0.000 to 0.000] | 5.130 [0.000 to 36.490] | 0.000 [0.000 to 0.000]
  WEEK12, EOI+5MIN: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+5MIN | 20.740 [20.500 to 20.980] |  | 66.540 [54.240 to 78.840] | 150.260 [105.080 to 157.210] | 98.041 [98.041 to 98.041]
  WEEK12, EOI+15MIN: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+15MIN | 20.720 [18.620 to 22.820] |  | 47.080 [37.990 to 56.170] | 132.160 [69.800 to 162.590] | 86.184 [86.184 to 86.184]
  WEEK12, EOI+30MIN: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+30MIN | 16.215 [13.430 to 19.000] |  | 41.385 [40.220 to 42.550] | 111.920 [59.310 to 125.540] | 85.491 [85.491 to 85.491]
  WEEK12, EOI+45MIN: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+45MIN | 11.150 [8.620 to 13.680] |  | 29.580 [26.990 to 32.170] | 89.030 [46.410 to 122.500] | 78.505 [78.505 to 78.505]
  WEEK12, EOI+1HR: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+1HR | 5.325 [0.000 to 10.650] |  | 24.850 [23.830 to 25.870] | 72.730 [36.330 to 118.150] | 61.492 [61.492 to 61.492]
  WEEK12, EOI+2HR: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+2HR | 3.205 [0.000 to 6.410] |  | 13.405 [11.900 to 14.910] | 64.050 [18.220 to 97.980] | 38.384 [38.384 to 38.384]
  WEEK12, EOI+4HR: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12, EOI+4HR | 0.000 [0.000 to 0.000] |  | 2.650 [0.000 to 5.300] | 19.080 [7.760 to 46.580] | 28.923 [28.923 to 28.923]
  WEEK12, EOI+8HR: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  WEEK12, EOI+8HR |  |  |  | 20.940 [20.940 to 20.940] |
  WEEK12, EOI+24HR: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  WEEK12, EOI+24HR |  |  |  | 6.730 [6.730 to 6.730] |
  WEEK19, PREDOSE: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  WEEK19, PREDOSE | 0.000 [0.000 to 13.000] | 0.000 [0.000 to 0.000] |  |  |
  WEEK19, EOI+5MIN: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  WEEK19, EOI+5MIN | 19.000 [15.700 to 31.000] | 42.400 [42.400 to 42.400] |  |  |
  WEEK19, EOI+2HR: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  WEEK19, EOI+2HR | 5.280 [3.930 to 5.390] | 24.100 [24.100 to 24.100] |  |  |
  WEEK19, EOI+4HR: number analyzed (Participants) | 3 | 1 | 0 | 0 | 0
  WEEK19, EOI+4HR | 1.540 [0.849 to 2.870] | 18.800 [18.800 to 18.800] |  |  |
  WEEK19, EOI+8HR: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK19, EOI+8HR | 0.409 [0.409 to 0.409] |  |  |  |
  WEEK55, PREDOSE: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK55, PREDOSE | 0.000 [0.000 to 0.000] |  |  |  |
  WEEK55, EOI+5MIN: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK55, EOI+5MIN | 13.500 [13.500 to 13.500] |  |  |  |
  WEEK55, EOI+2HR: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK55, EOI+2HR | 5.510 [5.510 to 5.510] |  |  |  |

9. Secondary Outcome: Part 1A: Area Under the Concentration-time Curve (AUC0-tau) Following Administration of GSK3745417 Alone (Q1W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1 to 6, 9, 10, 12, 19
Population: Pharmacokinetic (PK) population. The number analyzed for each timepoint reflects the number of participants from the Overall PK population with a non-missing value at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanogram/ millilitre (h*ng/mL)
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis
Number analyzed (Participants) | 14 | 2 | 17 | 10 | 7
Hours*Nanogram/ millilitre (h*ng/mL)
  WEEK1 | 47.0402 (73.0706) | 425.3023 (189.7100) | 145.6088 (111.8033) | 246.7692 (132.0408) | 247.2823 (79.1154)
  WEEK2: number analyzed (Participants) | 14 | 2 | 16 | 9 | 6
  WEEK2 | 77.8444 (108.5440) | 173.6723 (38.7832) | 130.5975 (114.5345) | 297.4580 (137.6797) | 253.8358 (103.5394)
  WEEK3: number analyzed (Participants) | 14 | 2 | 15 | 8 | 5
  WEEK3 | 69.7018 (102.8510) | 63.1059 (377.1988) | 150.3281 (116.4078) | 272.8593 (127.8989) | 198.6138 (70.3728)
  WEEK4: number analyzed (Participants) | 13 | 2 | 15 | 9 | 6
  WEEK4 | 46.2111 (126.0831) | 338.2702 (96.4149) | 133.7003 (132.4949) | 318.5676 (115.5291) | 234.0111 (85.9781)
  WEEK5: number analyzed (Participants) | 11 | 2 | 12 | 7 | 5
  WEEK5 | 46.6175 (103.7140) | 285.9155 (118.7575) | 149.6756 (122.4637) | 304.3914 (139.3329) | 203.4746 (53.4979)
  WEEK6: number analyzed (Participants) | 12 | 0 | 8 | 5 | 4
  WEEK6 | 38.6047 (101.8073) |  | 138.8428 (132.3027) | 245.7313 (103.6711) | 175.7315 (63.3206)
  WEEK9: number analyzed (Participants) | 3 | 0 | 1 | 3 | 3
  WEEK9 | 18.8752 (55.5837) |  | 79.7311 (NA) — GCV is not estimable as only a single participant was analyzed. | 199.9995 (61.2526) | 216.6902 (91.1146)
  WEEK10: number analyzed (Participants) | 5 | 0 | 1 | 0 | 0
  WEEK10 | 39.0336 (35.7876) |  | 133.8118 (NA) — GCV is not estimable as only a single participant was analyzed. |  |
  WEEK12: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12 | 19.8179 (61.7906) |  | 84.7136 (35.4645) | 276.5512 (116.8407) | 255.0798 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK19 | 28.6164 (NA) — GCV is not estimable as only a single participant was analyzed. |  |  |  |

10. Secondary Outcome: Part 1A: Maximum Observed Concentration (Cmax) Following Administration of GSK3745417 Alone (Q1W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1 to 6, 9, 10, 12, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis
Number analyzed (Participants) | 14 | 2 | 17 | 10 | 7
ng/mL
  WEEK1 | 21.648 (44.920) | 39.421 (40.108) | 53.434 (38.959) | 115.067 (21.459) | 115.244 (24.732)
  WEEK2: number analyzed (Participants) | 14 | 2 | 16 | 9 | 6
  WEEK2 | 24.710 (33.028) | 19.922 (59.477) | 47.747 (66.571) | 114.148 (27.392) | 111.111 (31.847)
  WEEK3: number analyzed (Participants) | 14 | 2 | 15 | 8 | 5
  WEEK3 | 25.079 (47.896) | 6.152 (248.490) | 49.458 (38.252) | 112.085 (26.349) | 103.552 (24.989)
  WEEK4: number analyzed (Participants) | 13 | 2 | 15 | 9 | 6
  WEEK4 | 20.791 (57.142) | 27.442 (24.724) | 46.712 (50.725) | 118.978 (21.611) | 125.171 (30.301)
  WEEK5: number analyzed (Participants) | 11 | 2 | 12 | 7 | 5
  WEEK5 | 18.057 (42.913) | 20.669 (37.429) | 50.470 (34.755) | 116.290 (35.137) | 117.339 (20.709)
  WEEK6: number analyzed (Participants) | 12 | 0 | 8 | 5 | 4
  WEEK6 | 17.284 (38.137) |  | 51.851 (84.399) | 120.172 (25.810) | 111.399 (13.175)
  WEEK9: number analyzed (Participants) | 3 | 0 | 1 | 3 | 3
  WEEK9 | 19.956 (44.055) |  | 43.320 (NA) — GCV is not estimable as only a single participant was analyzed. | 119.378 (46.814) | 111.267 (25.162)
  WEEK10: number analyzed (Participants) | 5 | 0 | 1 | 0 | 0
  WEEK10 | 18.972 (61.730) |  | 72.100 (NA) — GCV is not estimable as only a single participant was analyzed. |  |
  WEEK12: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12 | 24.213 (8.391) |  | 128.974 (71.075) | 151.763 (34.837) | 116.269 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK19 | 15.700 (NA) — GCV is not estimable as only a single participant was analyzed. |  |  |  |

11. Secondary Outcome: Part 1A: Apparent Terminal Phase Half-life (t1/2) Following Administration of GSK3745417 Alone (Q1W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1 to 6, 9, 10, 12, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis
Number analyzed (Participants) | 14 | 2 | 17 | 10 | 7
Hours
  WEEK1 | 2.6641 (106.8910) | 9.5995 (28.9474) | 3.9070 (210.2296) | 1.3649 (73.8778) | 5.8372 (277.8089)
  WEEK2: number analyzed (Participants) | 14 | 2 | 16 | 9 | 6
  WEEK2 | 4.7658 (328.9786) | 19.3880 (469.4324) | 2.9851 (142.5006) | 1.9345 (128.5751) | 3.0618 (71.7607)
  WEEK3: number analyzed (Participants) | 13 | 2 | 15 | 8 | 5
  WEEK3 | 3.7449 (206.4953) | 2.6123 (174.1372) | 3.3057 (155.8241) | 1.6793 (100.7945) | 3.6785 (30.4604)
  WEEK4: number analyzed (Participants) | 13 | 2 | 15 | 9 | 6
  WEEK4 | 3.5628 (254.2437) | 3.2869 (68.0644) | 2.8734 (146.3490) | 2.1743 (110.6625) | 5.4240 (106.1862)
  WEEK5: number analyzed (Participants) | 11 | 2 | 12 | 7 | 5
  WEEK5 | 3.3936 (231.5664) | 4.2877 (51.4222) | 3.6380 (215.0417) | 2.0752 (137.0553) | 3.1800 (29.9556)
  WEEK6: number analyzed (Participants) | 12 | 0 | 8 | 5 | 4
  WEEK6 | 2.8077 (90.0579) |  | 3.4171 (154.7470) | 1.9482 (136.5929) | 3.1452 (31.5377)
  WEEK9: number analyzed (Participants) | 3 | 0 | 1 | 3 | 3
  WEEK9 | 0.8472 (46.5385) |  | 1.1755 (NA) — GCV is not estimable as only a single participant was analyzed. | 1.1873 (30.5239) | 1.5023 (73.2964)
  WEEK10: number analyzed (Participants) | 5 | 0 | 1 | 0 | 0
  WEEK10 | 1.7913 (68.2418) |  | 1.5753 (NA) — GCV is not estimable as only a single participant was analyzed. |  |
  WEEK12: number analyzed (Participants) | 2 | 0 | 2 | 3 | 1
  WEEK12 | 0.7582 (77.8995) |  | 0.8903 (52.3388) | 1.8997 (167.2107) | 1.9083 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  WEEK19 | 1.3160 (NA) — GCV is not estimable as only a single participant was analyzed. |  |  |  |

12. Secondary Outcome: Part 1A: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 Alone (Q3W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Pre-dose on W 1, 4, 7, 10, 13, 16, 19; EOI+5min/ 15min/ 30 min/ 45 min/1HR/ 2HR/ 4HR on W 1, 4, 7, 10, 13, 16, 19; EOI+8HR/ 24HR on W 1, 4, 7, 10, 13, 16
Population: as for outcome 9
Measure: Median (Full Range); unit: Nanogram/ millilitre (ng/mL)
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W)
Number analyzed (Participants) | 3 | 6
Nanogram/ millilitre (ng/mL)
  WEEK1, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK1, EOI+5MIN | 19.656 [17.655 to 25.572] | 68.092 [49.614 to 162.468]
  WEEK1, EOI+15MIN | 17.848 [16.170 to 23.631] | 59.686 [33.494 to 155.317]
  WEEK1, EOI+30MIN | 16.010 [14.343 to 19.921] | 48.956 [36.096 to 125.040]
  WEEK1, EOI+45MIN | 14.122 [13.289 to 18.092] | 41.514 [24.915 to 117.454]
  WEEK1, EOI+1HR | 12.503 [11.200 to 15.045] | 32.591 [19.755 to 94.943]
  WEEK1, EOI+2HR | 8.103 [7.523 to 9.174] | 14.133 [8.873 to 56.505]
  WEEK1, EOI+4HR | 4.324 [4.272 to 5.012] | 5.024 [1.507 to 14.038]
  WEEK1, EOI+8HR | 1.306 [0.895 to 1.365] | 0.867 [0.405 to 7.079]
  WEEK1, EOI+24HR | 0.213 [0.210 to 0.267] | 0.390 [0.101 to 3.568]
  WEEK4, PREDOSE: number analyzed (Participants) | 3 | 5
  WEEK4, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK4, EOI+5MIN: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+5MIN | 19.178 [15.501 to 29.510] | 79.138 [39.037 to 98.366]
  WEEK4, EOI+15MIN: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+15MIN | 19.738 [13.381 to 25.756] | 60.396 [40.734 to 78.122]
  WEEK4, EOI+30MIN: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+30MIN | 17.016 [11.846 to 23.782] | 42.864 [31.276 to 58.776]
  WEEK4, EOI+45MIN: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+45MIN | 15.065 [10.255 to 19.001] | 36.750 [21.772 to 42.049]
  WEEK4, EOI+1HR: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+1HR | 14.628 [8.744 to 16.928] | 31.770 [16.324 to 34.248]
  WEEK4, EOI+2HR: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+2HR | 9.483 [6.382 to 11.708] | 14.780 [4.748 to 16.674]
  WEEK4, EOI+4HR: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+4HR | 3.133 [2.251 to 6.454] | 2.769 [1.980 to 4.640]
  WEEK4, EOI+8HR: number analyzed (Participants) | 3 | 4
  WEEK4, EOI+8HR | 1.067 [0.573 to 2.210] | 0.712 [0.392 to 1.412]
  WEEK4, EOI+24HR: number analyzed (Participants) | 3 | 3
  WEEK4, EOI+24HR | 0.172 [0.000 to 0.415] | 0.162 [0.103 to 0.287]
  WEEK7, PREDOSE: number analyzed (Participants) | 2 | 4
  WEEK7, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK7, EOI+5MIN: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+5MIN | 17.996 [14.010 to 21.982] | 56.701 [39.881 to 79.572]
  WEEK7, EOI+15MIN: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+15MIN | 15.603 [12.060 to 19.145] | 51.354 [34.819 to 68.696]
  WEEK7, EOI+30MIN: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+30MIN | 16.050 [13.469 to 18.631] | 43.613 [28.577 to 50.756]
  WEEK7, EOI+45MIN: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+45MIN | 14.383 [12.296 to 16.469] | 34.381 [18.854 to 43.681]
  WEEK7, EOI+1HR: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+1HR | 13.182 [11.505 to 14.858] | 30.738 [20.794 to 43.870]
  WEEK7, EOI+2HR: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+2HR | 8.885 [8.539 to 9.230] | 17.308 [10.424 to 23.124]
  WEEK7, EOI+4HR: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+4HR | 4.126 [2.818 to 5.433] | 4.005 [2.532 to 12.401]
  WEEK7, EOI+8HR: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+8HR | 1.730 [1.065 to 2.394] | 0.978 [0.397 to 2.525]
  WEEK7, EOI+24HR: number analyzed (Participants) | 2 | 4
  WEEK7, EOI+24HR | 0.224 [0.109 to 0.339] | 0.249 [0.140 to 0.667]
  WEEK10, PREDOSE: number analyzed (Participants) | 2 | 3
  WEEK10, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.108]
  WEEK10, EOI+5MIN: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+5MIN | 16.300 [11.069 to 21.530] | 72.010 [44.858 to 94.105]
  WEEK10, EOI+15MIN: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+15MIN | 14.881 [10.665 to 19.097] | 59.605 [37.610 to 77.265]
  WEEK10, EOI+30MIN: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+30MIN | 14.029 [10.063 to 17.995] | 52.583 [31.784 to 60.159]
  WEEK10, EOI+45MIN: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+45MIN | 12.552 [9.074 to 16.029] | 53.366 [25.714 to 67.141]
  WEEK10, EOI+1HR: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+1HR | 10.926 [8.387 to 13.465] | 44.280 [21.319 to 62.502]
  WEEK10, EOI+2HR: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+2HR | 6.899 [6.278 to 7.519] | 29.161 [9.557 to 42.098]
  WEEK10, EOI+4HR: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+4HR | 3.349 [3.052 to 3.645] | 14.945 [2.206 to 23.259]
  WEEK10, EOI+8HR: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+8HR | 1.178 [0.823 to 1.533] | 2.970 [0.673 to 4.567]
  WEEK10, EOI+24HR: number analyzed (Participants) | 2 | 3
  WEEK10, EOI+24HR | 0.186 [0.128 to 0.243] | 0.667 [0.176 to 1.368]
  WEEK13, PREDOSE: number analyzed (Participants) | 1 | 2
  WEEK13, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK13, EOI+5MIN: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+5MIN | 11.616 [11.616 to 11.616] | 52.322 [38.977 to 65.666]
  WEEK13, EOI+15MIN: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+15MIN | 9.839 [9.839 to 9.839] | 54.481 [36.068 to 72.893]
  WEEK13, EOI+30MIN: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+30MIN | 8.136 [8.136 to 8.136] | 45.104 [31.641 to 58.567]
  WEEK13, EOI+45MIN: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+45MIN | 6.717 [6.717 to 6.717] | 42.186 [26.765 to 57.606]
  WEEK13, EOI+1HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+1HR | 6.132 [6.132 to 6.132] | 39.095 [25.038 to 53.152]
  WEEK13, EOI+2HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+2HR | 3.484 [3.484 to 3.484] | 25.151 [14.376 to 35.925]
  WEEK13, EOI+4HR: number analyzed (Participants) | 0 | 2
  WEEK13, EOI+4HR |  | 15.093 [7.481 to 22.704]
  WEEK13, EOI+8HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+8HR | 0.380 [0.380 to 0.380] | 5.522 [2.244 to 8.799]
  WEEK13, EOI+24HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+24HR | 0.000 [0.000 to 0.000] | 1.165 [0.540 to 1.790]
  WEEK16, PREDOSE: number analyzed (Participants) | 2 | 2
  WEEK16, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK16, EOI+5MIN: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+5MIN | 20.721 [16.660 to 24.781] | 52.777 [51.400 to 54.153]
  WEEK16, EOI+15MIN: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+15MIN | 18.115 [14.726 to 21.504] | 37.137 [36.800 to 37.474]
  WEEK16, EOI+30MIN: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+30MIN | 16.677 [14.130 to 19.224] | 25.695 [25.100 to 26.290]
  WEEK16, EOI+45MIN: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+45MIN | 14.784 [13.002 to 16.565] | 25.281 [18.700 to 31.861]
  WEEK16, EOI+1HR: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+1HR | 12.920 [12.095 to 13.744] | 18.798 [15.400 to 22.195]
  WEEK16, EOI+2HR: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+2HR | 9.099 [7.608 to 10.590] | 13.221 [5.540 to 20.902]
  WEEK16, EOI+4HR: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+4HR | 5.529 [4.391 to 6.667] | 5.104 [1.410 to 8.798]
  WEEK16, EOI+8HR: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+8HR | 1.455 [0.388 to 2.521] | 1.806 [0.230 to 3.382]
  WEEK16, EOI+24HR: number analyzed (Participants) | 2 | 2
  WEEK16, EOI+24HR | 0.284 [0.113 to 0.455] | 0.297 [0.000 to 0.594]
  WEEK19, PREDOSE: number analyzed (Participants) | 1 | 1
  WEEK19, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK19, EOI+5MIN: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+5MIN | 24.762 [24.762 to 24.762] | 48.719 [48.719 to 48.719]
  WEEK19, EOI+15MIN: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+15MIN | 20.382 [20.382 to 20.382] | 41.813 [41.813 to 41.813]
  WEEK19, EOI+30MIN: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+30MIN | 19.166 [19.166 to 19.166] | 33.774 [33.774 to 33.774]
  WEEK19, EOI+45MIN: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+45MIN | 15.938 [15.938 to 15.938] | 28.790 [28.790 to 28.790]
  WEEK19, EOI+1HR: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+1HR | 13.778 [13.778 to 13.778] | 22.454 [22.454 to 22.454]
  WEEK19, EOI+2HR: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+2HR | 7.581 [7.581 to 7.581] | 21.388 [21.388 to 21.388]
  WEEK19, EOI+4HR: number analyzed (Participants) | 1 | 1
  WEEK19, EOI+4HR | 4.616 [4.616 to 4.616] | 10.894 [10.894 to 10.894]

13. Secondary Outcome: Part 1A: AUC(0-tau) Following Administration of GSK3745417 Alone (Q3W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1, 4, 7, 10, 13, 16, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*Nanogram/ millilitre (h*ng/mL)
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W)
Number analyzed (Participants) | 3 | 5
Hours*Nanogram/ millilitre (h*ng/mL)
  WEEK1 | 113.1657 (7.8510) | 145.2959 (49.6241)
  WEEK4: number analyzed (Participants) | 3 | 4
  WEEK4 | 87.6701 (97.5597) | 120.1116 (37.5649)
  WEEK7: number analyzed (Participants) | 2 | 4
  WEEK7 | 108.6757 (46.0604) | 160.3952 (60.7743)
  WEEK10: number analyzed (Participants) | 2 | 3
  WEEK10 | 55.1481 (20.7267) | 227.9506 (144.4144)
  WEEK13: number analyzed (Participants) | 1 | 2
  WEEK13 | 24.5659 (NA) — GCV is not estimable as only a single participant was analyzed. | 262.4978 (16.2226)
  WEEK16: number analyzed (Participants) | 2 | 2
  WEEK16 | 80.1101 (3.0157) | 96.6895 (103.2832)
  WEEK19: number analyzed (Participants) | 1 | 0
  WEEK19 | 47.0437 (NA) — GCV is not estimable as only a single participant was analyzed. |

14. Secondary Outcome: Part 1A: Cmax Following Administration of GSK3745417 Alone (Q3W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1, 4, 7, 10, 13, 16, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W)
Number analyzed (Participants) | 3 | 5
ng/mL
  WEEK1 | 20.703 (19.236) | 66.892 (24.171)
  WEEK4: number analyzed (Participants) | 3 | 4
  WEEK4 | 20.823 (33.402) | 79.308 (21.611)
  WEEK7: number analyzed (Participants) | 2 | 4
  WEEK7 | 17.549 (32.677) | 56.320 (30.480)
  WEEK10: number analyzed (Participants) | 2 | 3
  WEEK10 | 15.437 (49.771) | 67.238 (38.878)
  WEEK13: number analyzed (Participants) | 1 | 3
  WEEK13 | 11.616 (NA) — GCV is not estimable as only a single participant was analyzed. | 53.302 (46.526)
  WEEK16: number analyzed (Participants) | 2 | 2
  WEEK16 | 20.319 (28.639) | 52.759 (3.691)
  WEEK19: number analyzed (Participants) | 1 | 0
  WEEK19 | 24.762 (NA) — GCV is not estimable as only a single participant was analyzed. |

15. Secondary Outcome: Part 1A: T1/2 Following Administration of GSK3745417 Alone (Q3W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 alone.
Time Frame: Week 1, 4, 7, 10, 13, 16, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W)
Number analyzed (Participants) | 3 | 5
Hours
  WEEK1 | 3.3703 (8.6696) | 3.3373 (26.7810)
  WEEK4: number analyzed (Participants) | 3 | 4
  WEEK4 | 3.0907 (64.7708) | 3.2810 (97.7614)
  WEEK7: number analyzed (Participants) | 2 | 4
  WEEK7 | 4.3622 (8.6103) | 7.5933 (703.4471)
  WEEK10: number analyzed (Participants) | 2 | 3
  WEEK10 | 3.8978 (37.0772) | 4.0823 (26.7208)
  WEEK13: number analyzed (Participants) | 1 | 2
  WEEK13 | 1.6765 (NA) — GCV is not estimable as only a single participant was analyzed. | 4.7440 (42.2168)
  WEEK16: number analyzed (Participants) | 2 | 2
  WEEK16 | 3.5409 (35.5513) | 2.3492 (146.8761)
  WEEK19: number analyzed (Participants) | 1 | 0
  WEEK19 | 1.4041 (NA) — GCV is not estimable as only a single participant was analyzed. |

16. Secondary Outcome: Part 2A: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3745417 in combination with dostarlimab.
Time Frame: Pre-dose,EOI+5min/2HR/4HR on W 1 to 5, 7, 10, 13, 19, 37, 55; EOI+15min/ 30min/ 45 min/ 1HR on W 1, 4, 7; EOI+8HR on W 1 to 5, 7, 10, 13, 19; EOI+24HR on W 1 to 5, 7, 10
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 10
ng/mL
  WEEK1, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK1, EOI+5MIN | 26.350 [14.300 to 28.800] | 54.750 [26.600 to 86.600]
  WEEK1, EOI+15MIN | 23.150 [11.900 to 23.700] | 50.500 [21.400 to 76.400]
  WEEK1, EOI+30MIN | 20.450 [19.800 to 21.300] | 43.600 [19.400 to 76.100]
  WEEK1, EOI+45MIN | 17.550 [17.000 to 18.600] | 39.600 [14.200 to 68.800]
  WEEK1, EOI+1HR | 18.050 [15.600 to 22.300] | 34.800 [12.100 to 67.500]
  WEEK1, EOI+2HR | 12.400 [9.520 to 14.800] | 25.550 [3.630 to 55.000]
  WEEK1, EOI+4HR | 7.735 [5.360 to 9.620] | 14.650 [0.810 to 44.100]
  WEEK1, EOI+8HR: number analyzed (Participants) | 3 | 10
  WEEK1, EOI+8HR | 2.580 [0.631 to 3.920] | 5.880 [0.158 to 17.900]
  WEEK1, EOI+24HR | 0.390 [0.178 to 0.764] | 1.007 [0.000 to 3.710]
  WEEK2, PREDOSE: number analyzed (Participants) | 4 | 8
  WEEK2, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.165]
  WEEK2, EOI+5MIN: number analyzed (Participants) | 4 | 6
  WEEK2, EOI+5MIN | 19.250 [10.200 to 26.200] | 50.300 [31.300 to 91.400]
  WEEK2, EOI+2HR: number analyzed (Participants) | 4 | 8
  WEEK2, EOI+2HR | 14.900 [9.400 to 16.000] | 25.550 [8.600 to 57.300]
  WEEK2, EOI+4HR: number analyzed (Participants) | 4 | 7
  WEEK2, EOI+4HR | 10.105 [4.480 to 11.400] | 15.100 [1.840 to 40.000]
  WEEK2, EOI+8HR: number analyzed (Participants) | 4 | 5
  WEEK2, EOI+8HR | 5.105 [1.390 to 8.460] | 9.830 [2.060 to 21.900]
  WEEK2, EOI+24HR: number analyzed (Participants) | 0 | 2
  WEEK2, EOI+24HR |  | 3.915 [3.460 to 4.370]
  WEEK3, PREDOSE: number analyzed (Participants) | 3 | 8
  WEEK3, PREDOSE | 0.000 [0.000 to 0.211] | 0.000 [0.000 to 0.170]
  WEEK3, EOI+5MIN: number analyzed (Participants) | 2 | 7
  WEEK3, EOI+5MIN | 22.550 [20.900 to 24.200] | 49.700 [32.900 to 58.700]
  WEEK3, EOI+2HR: number analyzed (Participants) | 3 | 8
  WEEK3, EOI+2HR | 17.600 [10.200 to 18.200] | 25.300 [6.700 to 41.800]
  WEEK3, EOI+4HR: number analyzed (Participants) | 3 | 8
  WEEK3, EOI+4HR | 12.800 [5.930 to 14.200] | 14.000 [1.300 to 31.800]
  WEEK3, EOI+8HR: number analyzed (Participants) | 3 | 6
  WEEK3, EOI+8HR | 6.470 [2.770 to 10.200] | 6.535 [2.160 to 15.000]
  WEEK3, EOI+24HR: number analyzed (Participants) | 0 | 2
  WEEK3, EOI+24HR |  | 2.550 [2.040 to 3.060]
  WEEK4, PREDOSE: number analyzed (Participants) | 4 | 6
  WEEK4, PREDOSE | 0.000 [0.000 to 1.160] | 0.000 [0.000 to 0.000]
  WEEK4, EOI+5MIN: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+5MIN | 27.950 [19.200 to 45.700] | 39.400 [27.400 to 67.300]
  WEEK4, EOI+15MIN: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+15MIN | 24.950 [19.800 to 29.500] | 35.550 [23.800 to 55.300]
  WEEK4, EOI+30MIN: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+30MIN | 25.800 [16.300 to 31.300] | 31.100 [18.400 to 49.000]
  WEEK4, EOI+45MIN: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+45MIN | 21.150 [17.300 to 25.100] | 27.600 [13.700 to 43.000]
  WEEK4, EOI+1HR: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+1HR | 23.850 [16.300 to 24.700] | 25.650 [9.860 to 34.000]
  WEEK4, EOI+2HR: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+2HR | 18.100 [12.600 to 21.800] | 19.700 [3.840 to 21.700]
  WEEK4, EOI+4HR: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+4HR | 8.610 [7.750 to 17.700] | 10.300 [0.867 to 13.600]
  WEEK4, EOI+8HR: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+8HR | 4.275 [1.140 to 14.100] | 3.125 [0.256 to 6.470]
  WEEK4, EOI+24HR: number analyzed (Participants) | 4 | 6
  WEEK4, EOI+24HR | 0.675 [0.314 to 10.000] | 0.677 [0.000 to 1.040]
  WEEK5, PREDOSE: number analyzed (Participants) | 2 | 8
  WEEK5, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK5, EOI+5MIN: number analyzed (Participants) | 1 | 8
  WEEK5, EOI+5MIN | 16.300 [16.300 to 16.300] | 45.250 [34.900 to 58.100]
  WEEK5, EOI+2HR: number analyzed (Participants) | 2 | 8
  WEEK5, EOI+2HR | 10.375 [9.250 to 11.500] | 19.050 [9.380 to 23.900]
  WEEK5, EOI+4HR: number analyzed (Participants) | 2 | 8
  WEEK5, EOI+4HR | 5.670 [3.820 to 7.520] | 8.720 [2.160 to 17.200]
  WEEK5, EOI+8HR: number analyzed (Participants) | 2 | 7
  WEEK5, EOI+8HR | 2.484 [0.938 to 4.030] | 3.130 [0.937 to 14.300]
  WEEK5, EOI+24HR: number analyzed (Participants) | 0 | 2
  WEEK5, EOI+24HR |  | 0.719 [0.237 to 1.200]
  WEEK7, PREDOSE: number analyzed (Participants) | 1 | 6
  WEEK7, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 43.000]
  WEEK7, EOI+5MIN: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+5MIN | 19.600 [19.600 to 19.600] | 45.950 [38.600 to 79.500]
  WEEK7, EOI+15MIN: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+15MIN | 19.200 [19.200 to 19.200] | 40.650 [28.500 to 74.100]
  WEEK7, EOI+30MIN: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+30MIN | 15.000 [15.000 to 15.000] | 36.750 [24.900 to 66.700]
  WEEK7, EOI+45MIN: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+45MIN | 12.000 [12.000 to 12.000] | 32.900 [16.800 to 61.400]
  WEEK7, EOI+1HR: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+1HR | 10.200 [10.200 to 10.200] | 29.500 [11.500 to 60.900]
  WEEK7, EOI+2HR: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+2HR | 6.990 [6.990 to 6.990] | 18.400 [4.610 to 55.400]
  WEEK7, EOI+4HR: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+4HR | 3.090 [3.090 to 3.090] | 8.515 [0.920 to 34.900]
  WEEK7, EOI+8HR: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+8HR | 0.463 [0.463 to 0.463] | 2.340 [0.294 to 11.100]
  WEEK7, EOI+24HR: number analyzed (Participants) | 1 | 6
  WEEK7, EOI+24HR | 0.000 [0.000 to 0.000] | 0.528 [0.000 to 3.420]
  WEEK10, PREDOSE: number analyzed (Participants) | 1 | 6
  WEEK10, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK10, EOI+5MIN: number analyzed (Participants) | 1 | 6
  WEEK10, EOI+5MIN | 38.000 [38.000 to 38.000] | 49.700 [39.200 to 57.800]
  WEEK10, EOI+2HR: number analyzed (Participants) | 1 | 6
  WEEK10, EOI+2HR | 9.940 [9.940 to 9.940] | 17.550 [5.950 to 25.800]
  WEEK10, EOI+4HR: number analyzed (Participants) | 1 | 5
  WEEK10, EOI+4HR | 4.570 [4.570 to 4.570] | 6.710 [1.340 to 17.300]
  WEEK10, EOI+8HR: number analyzed (Participants) | 1 | 4
  WEEK10, EOI+8HR | 0.782 [0.782 to 0.782] | 4.840 [1.300 to 8.860]
  WEEK10, EOI+24HR: number analyzed (Participants) | 0 | 1
  WEEK10, EOI+24HR |  | 0.250 [0.250 to 0.250]
  WEEK13, PREDOSE: number analyzed (Participants) | 1 | 6
  WEEK13, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK13, EOI+5MIN: number analyzed (Participants) | 1 | 6
  WEEK13, EOI+5MIN | 22.100 [22.100 to 22.100] | 49.950 [42.300 to 58.100]
  WEEK13, EOI+2HR: number analyzed (Participants) | 1 | 6
  WEEK13, EOI+2HR | 9.220 [9.220 to 9.220] | 22.900 [3.310 to 45.500]
  WEEK13, EOI+4HR: number analyzed (Participants) | 1 | 6
  WEEK13, EOI+4HR | 5.110 [5.110 to 5.110] | 10.120 [0.627 to 20.800]
  WEEK13, EOI+8HR: number analyzed (Participants) | 1 | 4
  WEEK13, EOI+8HR | 1.140 [1.140 to 1.140] | 4.825 [3.780 to 12.100]
  WEEK19, PREDOSE: number analyzed (Participants) | 0 | 3
  WEEK19, PREDOSE |  | 0.000 [0.000 to 0.961]
  WEEK19, EOI+5MIN: number analyzed (Participants) | 0 | 3
  WEEK19, EOI+5MIN |  | 44.700 [42.900 to 64.000]
  WEEK19, EOI+2HR: number analyzed (Participants) | 0 | 3
  WEEK19, EOI+2HR |  | 17.400 [4.830 to 38.000]
  WEEK19, EOI+4HR: number analyzed (Participants) | 0 | 3
  WEEK19, EOI+4HR |  | 6.090 [0.678 to 34.700]
  WEEK19, EOI+8HR: number analyzed (Participants) | 0 | 1
  WEEK19, EOI+8HR |  | 21.800 [21.800 to 21.800]
  WEEK37, PREDOSE: number analyzed (Participants) | 0 | 1
  WEEK37, PREDOSE |  | 0.000 [0.000 to 0.000]
  WEEK37, EOI+5MIN: number analyzed (Participants) | 0 | 1
  WEEK37, EOI+5MIN |  | 51.400 [51.400 to 51.400]
  WEEK37, EOI+2HR: number analyzed (Participants) | 0 | 1
  WEEK37, EOI+2HR |  | 16.100 [16.100 to 16.100]
  WEEK37, EOI+4HR: number analyzed (Participants) | 0 | 1
  WEEK37, EOI+4HR |  | 6.150 [6.150 to 6.150]
  WEEK55, PREDOSE: number analyzed (Participants) | 0 | 1
  WEEK55, PREDOSE |  | 0.000 [0.000 to 0.000]
  WEEK55, EOI+5MIN: number analyzed (Participants) | 0 | 1
  WEEK55, EOI+5MIN |  | 123.000 [123.000 to 123.000]
  WEEK55, EOI+2HR: number analyzed (Participants) | 0 | 1
  WEEK55, EOI+2HR |  | 10.600 [10.600 to 10.600]
  WEEK55, EOI+4HR: number analyzed (Participants) | 0 | 1
  WEEK55, EOI+4HR |  | 3.310 [3.310 to 3.310]

17. Secondary Outcome: Part 2A: AUC(0-tau) Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Week 1 to 5, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 9
h*ng/mL
  WEEK1 | 105.7925 (37.9802) | 216.5303 (118.8420)
  WEEK2: number analyzed (Participants) | 4 | 7
  WEEK2 | 271.1541 (167.9069) | 471.1217 (96.1181)
  WEEK3: number analyzed (Participants) | 3 | 8
  WEEK3 | 326.3424 (105.6259) | 310.4697 (81.1473)
  WEEK4: number analyzed (Participants) | 4 | 6
  WEEK4 | 216.7790 (129.0498) | 130.8498 (76.6372)
  WEEK5: number analyzed (Participants) | 1 | 7
  WEEK5 | 93.7275 (NA) — GCV is not estimable as only a single participant was analyzed. | 128.9958 (39.4126)
  WEEK7: number analyzed (Participants) | 1 | 6
  WEEK7 | 43.3152 (NA) — GCV is not estimable as only a single participant was analyzed. | 130.9849 (80.5132)
  WEEK10: number analyzed (Participants) | 1 | 3
  WEEK10 | 69.6510 (NA) — GCV is not estimable as only a single participant was analyzed. | 122.3525 (31.6306)
  WEEK13: number analyzed (Participants) | 1 | 4
  WEEK13 | 87.5461 (NA) — GCV is not estimable as only a single participant was analyzed. | 171.3085 (31.4407)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 476.8171 (NA) — GCV is not estimable as only a single participant was analyzed.

18. Secondary Outcome: Part 2A: Cmax Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Week 1 to 5, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 9
ng/mL
  WEEK1 | 25.829 (11.287) | 51.212 (31.808)
  WEEK2: number analyzed (Participants) | 4 | 7
  WEEK2 | 17.709 (44.248) | 40.056 (72.883)
  WEEK3: number analyzed (Participants) | 3 | 8
  WEEK3 | 20.725 (16.041) | 44.277 (29.284)
  WEEK4: number analyzed (Participants) | 4 | 6
  WEEK4 | 29.271 (35.456) | 41.366 (31.911)
  WEEK5: number analyzed (Participants) | 1 | 7
  WEEK5 | 16.300 (NA) — GCV is not estimable as only a single participant was analyzed. | 42.791 (19.418)
  WEEK7: number analyzed (Participants) | 1 | 6
  WEEK7 | 19.600 (NA) — GCV is not estimable as only a single participant was analyzed. | 49.347 (27.385)
  WEEK10: number analyzed (Participants) | 1 | 3
  WEEK10 | 38.000 (NA) — GCV is not estimable as only a single participant was analyzed. | 51.623 (17.632)
  WEEK13: number analyzed (Participants) | 1 | 4
  WEEK13 | 22.100 (NA) — GCV is not estimable as only a single participant was analyzed. | 50.660 (10.597)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 42.900 (NA) — GCV is not estimable as only a single participant was analyzed.

19. Secondary Outcome: Part 2A: T1/2 Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Week 1 to 5, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 4 | 9
Hours
  WEEK1 | 4.9496 (25.3441) | 6.6082 (97.7169)
  WEEK2: number analyzed (Participants) | 4 | 7
  WEEK2 | 5.4788 (163.2744) | 3.2754 (147.9302)
  WEEK3: number analyzed (Participants) | 3 | 8
  WEEK3 | 8.0669 (323.3053) | 2.3642 (72.3718)
  WEEK4: number analyzed (Participants) | 4 | 6
  WEEK4 | 9.9205 (148.2505) | 3.7841 (83.5863)
  WEEK5: number analyzed (Participants) | 1 | 7
  WEEK5 | 3.8954 (NA) — GCV is not estimable as only a single participant was analyzed. | 2.5329 (39.3756)
  WEEK7: number analyzed (Participants) | 1 | 6
  WEEK7 | 1.7032 (NA) — GCV is not estimable as only a single participant was analyzed. | 5.5454 (43.6477)
  WEEK10: number analyzed (Participants) | 1 | 3
  WEEK10 | 1.8660 (NA) — GCV is not estimable as only a single participant was analyzed. | 2.5380 (40.5521)
  WEEK13: number analyzed (Participants) | 1 | 4
  WEEK13 | 2.2804 (NA) — GCV is not estimable as only a single participant was analyzed. | 2.3912 (21.7772)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 6.7964 (NA) — GCV is not estimable as only a single participant was analyzed.

20. Secondary Outcome: Part 2A: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 in Combination With Dostarlimab (Imaging Q1W)
Description: as for outcome 16
Time Frame: Pre-dose and EOI+5min/ 2HR/ 4HR on W 1, 2, 5, 6, 8, 11, 14, 20, 38; EOI+15min/ 30min/ 45min/ 1HR/ 6HR on W 1 and 8; EOI+8HR in W 1, 2, 5, 6, 8; EOI+24HR on W 1, 2, 5, 8.
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 3 | 1
ng/mL
  WEEK1, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK1, EOI+5MIN: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+5MIN | 19.600 [9.060 to 20.300] |
  WEEK1, EOI+15MIN: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+15MIN | 19.000 [17.400 to 19.200] |
  WEEK1, EOI+30MIN: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+30MIN | 15.900 [14.700 to 18.100] |
  WEEK1, EOI+45MIN: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+45MIN | 13.700 [12.000 to 16.300] |
  WEEK1, EOI+1HR: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+1HR | 11.700 [10.500 to 14.100] |
  WEEK1, EOI+2HR: number analyzed (Participants) | 2 | 0
  WEEK1, EOI+2HR | 8.360 [6.750 to 9.970] |
  WEEK1, EOI+4HR: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+4HR | 2.290 [2.000 to 5.660] |
  WEEK1, EOI+6HR: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+6HR | 0.838 [0.765 to 2.980] |
  WEEK1, EOI+8HR: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+8HR | 0.374 [0.363 to 1.640] |
  WEEK1, EOI+24HR: number analyzed (Participants) | 3 | 0
  WEEK1, EOI+24HR | 0.204 [0.000 to 0.329] |
  WEEK2, PREDOSE | 0.000 [0.000 to 0.000] | 0.464 [0.464 to 0.464]
  WEEK2, EOI+5MIN | 12.200 [8.600 to 18.300] | 18.700 [18.700 to 18.700]
  WEEK2, EOI+2HR | 5.930 [3.280 to 8.680] | 17.200 [17.200 to 17.200]
  WEEK2, EOI+4HR: number analyzed (Participants) | 3 | 0
  WEEK2, EOI+4HR | 2.140 [1.190 to 5.030] |
  WEEK2, EOI+8HR | 0.425 [0.208 to 1.960] | 16.300 [16.300 to 16.300]
  WEEK2, EOI+24HR | 0.000 [0.000 to 0.181] | 9.210 [9.210 to 9.210]
  WEEK5, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK5, EOI+5MIN | 14.100 [8.990 to 15.600] | 82.500 [82.500 to 82.500]
  WEEK5, EOI+2HR | 6.910 [6.570 to 9.940] | 29.800 [29.800 to 29.800]
  WEEK5, EOI+4HR | 3.750 [1.850 to 5.180] | 15.100 [15.100 to 15.100]
  WEEK5, EOI+8HR | 1.440 [0.444 to 1.600] | 5.740 [5.740 to 5.740]
  WEEK5, EOI+24HR | 0.144 [0.000 to 0.238] | 0.571 [0.571 to 0.571]
  WEEK6, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK6, EOI+5MIN | 17.400 [13.500 to 20.600] | 53.000 [53.000 to 53.000]
  WEEK6, EOI+2HR | 7.790 [5.620 to 7.840] | 27.300 [27.300 to 27.300]
  WEEK6, EOI+4HR | 3.430 [1.570 to 4.370] | 13.000 [13.000 to 13.000]
  WEEK6, EOI+8HR: number analyzed (Participants) | 2 | 1
  WEEK6, EOI+8HR | 1.500 [1.390 to 1.610] | 5.670 [5.670 to 5.670]
  WEEK8, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK8, EOI+5MIN | 18.100 [12.000 to 21.300] | 64.400 [64.400 to 64.400]
  WEEK8, EOI+15MIN | 17.400 [14.400 to 18.700] | 52.900 [52.900 to 52.900]
  WEEK8, EOI+30MIN | 14.200 [11.100 to 18.700] | 50.500 [50.500 to 50.500]
  WEEK8, EOI+45MIN | 11.700 [9.990 to 16.000] | 43.800 [43.800 to 43.800]
  WEEK8, EOI+1HR | 10.400 [8.660 to 14.800] | 40.000 [40.000 to 40.000]
  WEEK8, EOI+2HR | 6.300 [4.810 to 10.200] | 26.600 [26.600 to 26.600]
  WEEK8, EOI+4HR | 1.700 [1.560 to 5.570] | 11.900 [11.900 to 11.900]
  WEEK8, EOI+6HR | 1.040 [0.563 to 3.310] | 7.130 [7.130 to 7.130]
  WEEK8, EOI+8HR | 0.626 [0.269 to 2.160] | 5.170 [5.170 to 5.170]
  WEEK8, EOI+24HR | 0.000 [0.000 to 0.309] | 0.548 [0.548 to 0.548]
  WEEK11, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK11, EOI+5MIN | 15.100 [8.820 to 20.800] | 68.300 [68.300 to 68.300]
  WEEK11, EOI+2HR | 8.790 [3.990 to 10.800] | 28.800 [28.800 to 28.800]
  WEEK11, EOI+4HR | 4.910 [1.310 to 6.530] | 14.300 [14.300 to 14.300]
  WEEK14, PREDOSE: number analyzed (Participants) | 2 | 1
  WEEK14, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK14, EOI+5MIN: number analyzed (Participants) | 2 | 1
  WEEK14, EOI+5MIN | 10.990 [5.480 to 16.500] | 56.800 [56.800 to 56.800]
  WEEK14, EOI+2HR: number analyzed (Participants) | 2 | 1
  WEEK14, EOI+2HR | 7.010 [4.800 to 9.220] | 12.500 [12.500 to 12.500]
  WEEK14, EOI+4HR: number analyzed (Participants) | 2 | 1
  WEEK14, EOI+4HR | 2.515 [1.730 to 3.300] | 6.850 [6.850 to 6.850]
  WEEK20, PREDOSE: number analyzed (Participants) | 1 | 0
  WEEK20, PREDOSE | 0.000 [0.000 to 0.000] |
  WEEK20, EOI+5MIN: number analyzed (Participants) | 1 | 0
  WEEK20, EOI+5MIN | 19.100 [19.100 to 19.100] |
  WEEK20, EOI+2HR: number analyzed (Participants) | 1 | 0
  WEEK20, EOI+2HR | 11.600 [11.600 to 11.600] |
  WEEK20, EOI+4HR: number analyzed (Participants) | 1 | 0
  WEEK20, EOI+4HR | 6.390 [6.390 to 6.390] |
  WEEK38, PREDOSE: number analyzed (Participants) | 1 | 0
  WEEK38, PREDOSE | 0.000 [0.000 to 0.000] |
  WEEK38, EOI+5MIN: number analyzed (Participants) | 1 | 0
  WEEK38, EOI+5MIN | 19.300 [19.300 to 19.300] |
  WEEK38, EOI+2HR: number analyzed (Participants) | 1 | 0
  WEEK38, EOI+2HR | 6.800 [6.800 to 6.800] |
  WEEK38, EOI+4HR: number analyzed (Participants) | 1 | 0
  WEEK38, EOI+4HR | 2.030 [2.030 to 2.030] |

21. Secondary Outcome: Part 2A: AUC(0-tau) Following Administration of GSK3745417 in Combination With Dostarlimab (Imaging Q1W)
Description: as for outcome 16
Time Frame: Week 1, 2, 5, 6, 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 3 | 1
h*ng/mL
  WEEK1: number analyzed (Participants) | 3 | 0
  WEEK1 | 61.7410 (41.6380) |
  WEEK2 | 35.1903 (67.6550) | 561.8580 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK5 | 50.7155 (51.4681) | 262.5058 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK6: number analyzed (Participants) | 2 | 1
  WEEK6 | 48.4490 (7.7001) | 163.2896 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK8 | 44.6483 (53.3204) | 187.0690 (NA) — GCV is not estimable as only a single participant was analyzed.

22. Secondary Outcome: Part 2A: Cmax Following Administration of GSK3745417 in Combination With Dostarlimab (Imaging Q1W)
Description: as for outcome 16
Time Frame: Week 1, 2, 5, 6, 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 3 | 1
ng/mL
  WEEK1: number analyzed (Participants) | 3 | 0
  WEEK1 | 19.695 (2.817) |
  WEEK2 | 12.429 (39.182) | 18.700 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK5 | 12.552 (29.984) | 82.500 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK6: number analyzed (Participants) | 2 | 1
  WEEK6 | 15.326 (18.090) | 53.000 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK8 | 18.860 (10.751) | 64.400 (NA) — GCV is not estimable as only a single participant was analyzed.

23. Secondary Outcome: Part 2A: T1/2 Following Administration of GSK3745417 in Combination With Dostarlimab (Imaging Q1W)
Description: as for outcome 16
Time Frame: Week 1, 2, 5, 6, 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 3 | 1
Hours
  WEEK1: number analyzed (Participants) | 3 | 0
  WEEK1 | 2.8013 (71.6405) |
  WEEK2 | 2.1751 (65.5517) | 22.0749 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK5 | 2.9851 (75.7387) | 4.4441 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK6: number analyzed (Participants) | 2 | 1
  WEEK6 | 2.2228 (0.3535) | 2.1489 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK8 | 2.1554 (97.4160) | 4.4423 (NA) — GCV is not estimable as only a single participant was analyzed.

24. Secondary Outcome: Part 2A: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Pre-dose on W 1, 4, 7, 10, 13, 19, 37, 55, 73, 91; EOI+5min/ 4HR on W 1, 4, 7, 10, 13, 19, 37, 55, 91; EOI+15min/ 30min/ 45min/ 1HR/ 6HR on W 1, 4, 7; EOI+2HR on W 1, 4, 7, 10, 13, 19, 37, 55, 73; EOI+8HR/24 HR on W 1, 4, 7, 10, 13, 19, 91
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 4 | 12
ng/mL
  WEEK1, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK1, EOI+5MIN | 23.100 [20.100 to 27.100] | 43.250 [25.200 to 78.700]
  WEEK1, EOI+15MIN | 20.550 [18.100 to 22.700] | 39.550 [20.300 to 61.700]
  WEEK1, EOI+30MIN | 16.600 [15.300 to 17.100] | 34.050 [15.900 to 56.500]
  WEEK1, EOI+45MIN | 13.100 [12.300 to 15.100] | 29.550 [12.000 to 49.100]
  WEEK1, EOI+1HR | 10.355 [9.300 to 13.000] | 26.550 [9.700 to 40.400]
  WEEK1, EOI+2HR | 4.260 [3.090 to 10.500] | 16.050 [2.400 to 30.000]
  WEEK1, EOI+4HR | 1.298 [0.514 to 4.550] | 6.055 [0.608 to 25.500]
  WEEK1, EOI+6HR | 0.512 [0.201 to 1.940] | 2.745 [0.280 to 18.500]
  WEEK1, EOI+8HR | 0.245 [0.167 to 0.952] | 1.160 [0.140 to 15.100]
  WEEK1, EOI+24HR | 0.000 [0.000 to 0.265] | 0.302 [0.000 to 6.660]
  WEEK4, PREDOSE: number analyzed (Participants) | 4 | 10
  WEEK4, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK4, EOI+5MIN: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+5MIN | 24.200 [22.700 to 26.000] | 42.400 [31.400 to 56.400]
  WEEK4, EOI+15MIN: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+15MIN | 20.800 [18.200 to 24.300] | 40.900 [25.200 to 50.200]
  WEEK4, EOI+30MIN: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+30MIN | 16.050 [13.700 to 18.700] | 34.700 [19.100 to 40.000]
  WEEK4, EOI+45MIN: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+45MIN | 12.800 [9.760 to 16.000] | 31.300 [15.300 to 38.800]
  WEEK4, EOI+1HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+1HR | 10.370 [6.680 to 17.000] | 28.200 [12.100 to 34.200]
  WEEK4, EOI+2HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+2HR | 3.905 [0.243 to 11.000] | 16.650 [5.230 to 25.500]
  WEEK4, EOI+4HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+4HR | 1.064 [0.237 to 4.090] | 6.095 [1.220 to 20.500]
  WEEK4, EOI+6HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+6HR | 0.355 [0.141 to 2.000] | 2.360 [0.471 to 14.800]
  WEEK4, EOI+8HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+8HR | 0.198 [0.114 to 1.110] | 1.141 [0.299 to 11.400]
  WEEK4, EOI+24HR: number analyzed (Participants) | 4 | 10
  WEEK4, EOI+24HR | 0.000 [0.000 to 0.266] | 0.221 [0.000 to 2.400]
  WEEK7, PREDOSE: number analyzed (Participants) | 3 | 7
  WEEK7, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 11.000]
  WEEK7, EOI+5MIN: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+5MIN | 21.400 [13.700 to 29.200] | 39.800 [28.900 to 52.700]
  WEEK7, EOI+15MIN: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+15MIN | 18.300 [14.800 to 31.800] | 34.300 [12.900 to 49.800]
  WEEK7, EOI+30MIN: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+30MIN | 14.500 [6.860 to 30.600] | 28.100 [6.610 to 40.600]
  WEEK7, EOI+45MIN: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+45MIN | 11.400 [6.430 to 24.100] | 26.400 [2.600 to 38.700]
  WEEK7, EOI+1HR: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+1HR | 9.080 [5.180 to 20.800] | 22.900 [0.464 to 32.400]
  WEEK7, EOI+2HR: number analyzed (Participants) | 3 | 6
  WEEK7, EOI+2HR | 4.130 [1.430 to 15.000] | 16.250 [7.220 to 25.000]
  WEEK7, EOI+4HR: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+4HR | 0.847 [0.223 to 5.630] | 6.820 [1.790 to 16.400]
  WEEK7, EOI+6HR: number analyzed (Participants) | 2 | 7
  WEEK7, EOI+6HR | 0.225 [0.122 to 0.328] | 3.610 [0.692 to 16.400]
  WEEK7, EOI+8HR: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+8HR | 0.137 [0.000 to 1.940] | 2.040 [0.310 to 9.710]
  WEEK7, EOI+24HR: number analyzed (Participants) | 3 | 7
  WEEK7, EOI+24HR | 0.000 [0.000 to 0.410] | 0.482 [0.114 to 5.340]
  WEEK10, PREDOSE: number analyzed (Participants) | 3 | 6
  WEEK10, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.159]
  WEEK10, EOI+5MIN: number analyzed (Participants) | 3 | 5
  WEEK10, EOI+5MIN | 22.900 [22.000 to 34.500] | 28.800 [24.100 to 47.500]
  WEEK10, EOI+2HR: number analyzed (Participants) | 3 | 6
  WEEK10, EOI+2HR | 4.270 [2.030 to 13.800] | 15.550 [8.030 to 25.500]
  WEEK10, EOI+4HR: number analyzed (Participants) | 3 | 6
  WEEK10, EOI+4HR | 1.080 [0.314 to 6.020] | 7.200 [2.740 to 14.600]
  WEEK10, EOI+8HR: number analyzed (Participants) | 2 | 4
  WEEK10, EOI+8HR | 0.094 [0.000 to 0.187] | 3.135 [0.750 to 6.320]
  WEEK10, EOI+24HR: number analyzed (Participants) | 0 | 2
  WEEK10, EOI+24HR |  | 1.015 [0.109 to 1.920]
  WEEK13, PREDOSE: number analyzed (Participants) | 3 | 3
  WEEK13, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK13, EOI+5MIN: number analyzed (Participants) | 3 | 2
  WEEK13, EOI+5MIN | 19.600 [17.400 to 20.700] | 51.350 [42.200 to 60.500]
  WEEK13, EOI+2HR: number analyzed (Participants) | 3 | 2
  WEEK13, EOI+2HR | 2.860 [1.330 to 9.930] | 25.000 [24.100 to 25.900]
  WEEK13, EOI+4HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+4HR | 5.870 [5.870 to 5.870] | 12.190 [9.380 to 15.000]
  WEEK13, EOI+8HR: number analyzed (Participants) | 1 | 2
  WEEK13, EOI+8HR | 0.399 [0.399 to 0.399] | 4.060 [2.990 to 5.130]
  WEEK13, EOI+24HR: number analyzed (Participants) | 0 | 2
  WEEK13, EOI+24HR |  | 1.227 [0.583 to 1.870]
  WEEK19, PREDOSE: number analyzed (Participants) | 2 | 2
  WEEK19, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK19, EOI+5MIN: number analyzed (Participants) | 2 | 2
  WEEK19, EOI+5MIN | 20.350 [17.400 to 23.300] | 85.950 [59.900 to 112.000]
  WEEK19, EOI+2HR: number analyzed (Participants) | 2 | 2
  WEEK19, EOI+2HR | 4.205 [3.290 to 5.120] | 43.200 [26.800 to 59.600]
  WEEK19, EOI+4HR: number analyzed (Participants) | 1 | 2
  WEEK19, EOI+4HR | 0.870 [0.870 to 0.870] | 23.600 [11.400 to 35.800]
  WEEK19, EOI+8HR: number analyzed (Participants) | 0 | 1
  WEEK19, EOI+8HR |  | 17.500 [17.500 to 17.500]
  WEEK19, EOI+24HR: number analyzed (Participants) | 0 | 1
  WEEK19, EOI+24HR |  | 3.490 [3.490 to 3.490]
  WEEK37, PREDOSE: number analyzed (Participants) | 1 | 1
  WEEK37, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK37, EOI+5MIN: number analyzed (Participants) | 1 | 0
  WEEK37, EOI+5MIN | 27.200 [27.200 to 27.200] |
  WEEK37, EOI+2HR: number analyzed (Participants) | 1 | 1
  WEEK37, EOI+2HR | 3.280 [3.280 to 3.280] | 20.100 [20.100 to 20.100]
  WEEK37, EOI+4HR: number analyzed (Participants) | 1 | 1
  WEEK37, EOI+4HR | 0.605 [0.605 to 0.605] | 7.430 [7.430 to 7.430]
  WEEK55, PREDOSE: number analyzed (Participants) | 1 | 1
  WEEK55, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  WEEK55, EOI+5MIN: number analyzed (Participants) | 1 | 0
  WEEK55, EOI+5MIN | 22.700 [22.700 to 22.700] |
  WEEK55, EOI+2HR: number analyzed (Participants) | 1 | 1
  WEEK55, EOI+2HR | 2.050 [2.050 to 2.050] | 17.300 [17.300 to 17.300]
  WEEK55, EOI+4HR: number analyzed (Participants) | 1 | 1
  WEEK55, EOI+4HR | 0.338 [0.338 to 0.338] | 8.660 [8.660 to 8.660]
  WEEK73, PREDOSE: number analyzed (Participants) | 1 | 0
  WEEK73, PREDOSE | 0.204 [0.204 to 0.204] |
  WEEK73, EOI+2HR: number analyzed (Participants) | 1 | 0
  WEEK73, EOI+2HR | 2.770 [2.770 to 2.770] |
  WEEK91, PREDOSE: number analyzed (Participants) | 1 | 0
  WEEK91, PREDOSE | 0.000 [0.000 to 0.000] |
  WEEK91, EOI+5MIN: number analyzed (Participants) | 1 | 0
  WEEK91, EOI+5MIN | 19.900 [19.900 to 19.900] |
  WEEK91, EOI+4HR: number analyzed (Participants) | 1 | 0
  WEEK91, EOI+4HR | 1.070 [1.070 to 1.070] |
  WEEK91, EOI+8HR: number analyzed (Participants) | 1 | 0
  WEEK91, EOI+8HR | 0.242 [0.242 to 0.242] |
  WEEK91, EOI+24HR: number analyzed (Participants) | 1 | 0
  WEEK91, EOI+24HR | 0.000 [0.000 to 0.000] |

25. Secondary Outcome: Part 2A: AUC(0-tau) Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Week 1, 4, 7, 10, 13, 19, 91
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 4 | 12
h*ng/mL
  WEEK1 | 41.2241 (46.8260) | 136.9391 (91.3047)
  WEEK4: number analyzed (Participants) | 4 | 9
  WEEK4 | 42.0297 (92.4823) | 110.3856 (83.9274)
  WEEK7: number analyzed (Participants) | 3 | 7
  WEEK7 | 44.0290 (208.4637) | 217.9598 (148.0574)
  WEEK10: number analyzed (Participants) | 3 | 3
  WEEK10 | 103.5186 (400.0481) | 283.2979 (364.4200)
  WEEK13: number analyzed (Participants) | 0 | 2
  WEEK13 |  | 189.3316 (16.9323)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 539.0039 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK91: number analyzed (Participants) | 1 | 0
  WEEK91 | 31.1811 (NA) — GCV is not estimable as only a single participant was analyzed. |

26. Secondary Outcome: Part 2A: Cmax Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Week 1, 4, 7, 10, 13, 19, 91
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 4 | 12
ng/mL
  WEEK1 | 23.184 (13.852) | 42.961 (26.296)
  WEEK4: number analyzed (Participants) | 4 | 10
  WEEK4 | 24.297 (5.545) | 42.936 (20.005)
  WEEK7: number analyzed (Participants) | 3 | 7
  WEEK7 | 23.179 (29.068) | 38.655 (20.087)
  WEEK10: number analyzed (Participants) | 3 | 3
  WEEK10 | 25.904 (25.290) | 29.947 (33.758)
  WEEK13: number analyzed (Participants) | 0 | 2
  WEEK13 |  | 50.528 (25.890)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 112.000 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK91: number analyzed (Participants) | 1 | 0
  WEEK91 | 19.900 (NA) — GCV is not estimable as only a single participant was analyzed. |

27. Secondary Outcome: Part 2A: T1/2 Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Week 1, 4, 7, 10, 13, 19, 91
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 4 | 12
Hours
  WEEK1 | 1.6491 (105.7556) | 4.5289 (65.1077)
  WEEK4: number analyzed (Participants) | 4 | 9
  WEEK4 | 1.7825 (64.9647) | 5.4869 (96.3549)
  WEEK7: number analyzed (Participants) | 3 | 7
  WEEK7 | 1.7101 (121.4103) | 10.1871 (122.2331)
  WEEK10: number analyzed (Participants) | 3 | 3
  WEEK10 | 1.1499 (54.3836) | 3.9067 (59.4336)
  WEEK13: number analyzed (Participants) | 0 | 2
  WEEK13 |  | 5.6356 (1.5314)
  WEEK19: number analyzed (Participants) | 0 | 1
  WEEK19 |  | 6.5557 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK91: number analyzed (Participants) | 1 | 0
  WEEK91 | 1.2513 (NA) — GCV is not estimable as only a single participant was analyzed. |

28. Secondary Outcome: Crossover Phase: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Pre-dose and EOI+5min/2HR/ 4HR/ 8HR on crossover W 1, 4, 7, 10, 13, 19; EOI+12HR/18HR on crossover W 4; EOI+15min/ 30 min/45 min/1HR/6HR/24HR on crossover W 1, 4, 7
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 1 | 4
ng/mL
  WEEK1 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 3
  WEEK1 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.639]
  WEEK1 CROSSOVER, EOI+5MIN | 28.900 [28.900 to 28.900] | 39.400 [23.600 to 65.500]
  WEEK1 CROSSOVER, EOI+15MIN | 22.800 [22.800 to 22.800] | 40.550 [32.700 to 68.300]
  WEEK1 CROSSOVER, EOI+30MIN: number analyzed (Participants) | 1 | 3
  WEEK1 CROSSOVER, EOI+30MIN | 18.600 [18.600 to 18.600] | 31.900 [28.800 to 38.600]
  WEEK1 CROSSOVER, EOI+45MIN | 17.300 [17.300 to 17.300] | 29.650 [25.900 to 47.300]
  WEEK1 CROSSOVER, EOI+1HR | 14.200 [14.200 to 14.200] | 27.000 [24.000 to 32.600]
  WEEK1 CROSSOVER, EOI+2HR | 10.300 [10.300 to 10.300] | 19.600 [8.430 to 26.300]
  WEEK1 CROSSOVER, EOI+4HR | 6.320 [6.320 to 6.320] | 12.025 [1.880 to 27.300]
  WEEK1 CROSSOVER, EOI+6HR | 4.780 [4.780 to 4.780] | 8.885 [0.740 to 14.500]
  WEEK1 CROSSOVER, EOI+8HR | 6.940 [6.940 to 6.940] | 2.835 [0.380 to 11.200]
  WEEK1 CROSSOVER, EOI+24HR | 3.780 [3.780 to 3.780] | 0.327 [0.000 to 5.920]
  WEEK4 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, PREDOSE | 8.340 [8.340 to 8.340] | 0.000 [0.000 to 0.155]
  WEEK4 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+5MIN | 14.200 [14.200 to 14.200] | 49.100 [39.100 to 50.000]
  WEEK4 CROSSOVER, EOI+15MIN: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+15MIN | 13.200 [13.200 to 13.200] | 45.100 [38.600 to 55.400]
  WEEK4 CROSSOVER, EOI+30MIN: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+30MIN | 16.100 [16.100 to 16.100] | 38.700 [35.900 to 40.800]
  WEEK4 CROSSOVER, EOI+45MIN: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+45MIN | 10.500 [10.500 to 10.500] | 38.000 [34.700 to 38.200]
  WEEK4 CROSSOVER, EOI+1HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+1HR | 10.200 [10.200 to 10.200] | 33.700 [30.600 to 34.400]
  WEEK4 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+2HR | 6.490 [6.490 to 6.490] | 23.200 [19.800 to 25.000]
  WEEK4 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+4HR | 6.330 [6.330 to 6.330] | 12.400 [6.890 to 15.000]
  WEEK4 CROSSOVER, EOI+6HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+6HR | 8.820 [8.820 to 8.820] | 5.740 [2.260 to 10.100]
  WEEK4 CROSSOVER, EOI+8HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+8HR | 4.760 [4.760 to 4.760] | 4.290 [1.140 to 9.530]
  WEEK4 CROSSOVER, EOI+12HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+12HR | 4.470 [4.470 to 4.470] | 1.560 [0.652 to 2.820]
  WEEK4 CROSSOVER, EOI+18HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+18HR | 10.600 [10.600 to 10.600] | 0.969 [0.431 to 1.760]
  WEEK4 CROSSOVER, EOI+24HR: number analyzed (Participants) | 1 | 3
  WEEK4 CROSSOVER, EOI+24HR | 2.180 [2.180 to 2.180] | 0.719 [0.366 to 1.400]
  WEEK7 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, PREDOSE | 3.320 [3.320 to 3.320] | 0.000 [0.000 to 0.000]
  WEEK7 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+5MIN | 25.000 [25.000 to 25.000] | 48.000 [35.600 to 60.400]
  WEEK7 CROSSOVER, EOI+15MIN: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+15MIN | 18.700 [18.700 to 18.700] | 40.750 [34.100 to 47.400]
  WEEK7 CROSSOVER, EOI+30MIN: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+30MIN | 20.500 [20.500 to 20.500] | 37.300 [29.100 to 45.500]
  WEEK7 CROSSOVER, EOI+45MIN: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+45MIN | 17.400 [17.400 to 17.400] | 34.450 [26.000 to 42.900]
  WEEK7 CROSSOVER, EOI+1HR: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+1HR | 16.100 [16.100 to 16.100] | 32.650 [24.700 to 40.600]
  WEEK7 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+2HR | 8.290 [8.290 to 8.290] | 23.500 [16.200 to 30.800]
  WEEK7 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+4HR | 7.130 [7.130 to 7.130] | 12.290 [9.080 to 15.500]
  WEEK7 CROSSOVER, EOI+6HR: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+6HR | 11.700 [11.700 to 11.700] | 6.350 [5.150 to 7.550]
  WEEK7 CROSSOVER, EOI+8HR: number analyzed (Participants) | 1 | 1
  WEEK7 CROSSOVER, EOI+8HR | 4.700 [4.700 to 4.700] | 4.740 [4.740 to 4.740]
  WEEK7 CROSSOVER, EOI+24HR: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER, EOI+24HR | 3.210 [3.210 to 3.210] | 0.822 [0.584 to 1.060]
  WEEK10 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000] | 0.085 [0.000 to 0.169]
  WEEK10 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER, EOI+5MIN | 10.700 [10.700 to 10.700] | 40.000 [33.300 to 46.700]
  WEEK10 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER, EOI+2HR | 3.400 [3.400 to 3.400] | 17.950 [15.100 to 20.800]
  WEEK10 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER, EOI+4HR | 2.300 [2.300 to 2.300] | 9.765 [9.130 to 10.400]
  WEEK10 CROSSOVER, EOI+8HR: number analyzed (Participants) | 0 | 2
  WEEK10 CROSSOVER, EOI+8HR |  | 3.665 [2.900 to 4.430]
  WEEK13 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 2
  WEEK13 CROSSOVER, PREDOSE | 3.970 [3.970 to 3.970] | 0.000 [0.000 to 0.000]
  WEEK13 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1 | 2
  WEEK13 CROSSOVER, EOI+5MIN | 22.700 [22.700 to 22.700] | 48.150 [30.000 to 66.300]
  WEEK13 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1 | 2
  WEEK13 CROSSOVER, EOI+2HR | 9.580 [9.580 to 9.580] | 29.650 [28.200 to 31.100]
  WEEK13 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1 | 2
  WEEK13 CROSSOVER, EOI+4HR | 5.140 [5.140 to 5.140] | 15.500 [14.900 to 16.100]
  WEEK13 CROSSOVER, EOI+8HR: number analyzed (Participants) | 0 | 1
  WEEK13 CROSSOVER, EOI+8HR |  | 6.070 [6.070 to 6.070]
  WEEK19 CROSSOVER, PREDOSE: number analyzed (Participants) | 1 | 2
  WEEK19 CROSSOVER, PREDOSE | 4.110 [4.110 to 4.110] | 0.362 [0.000 to 0.723]
  WEEK19 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1 | 2
  WEEK19 CROSSOVER, EOI+5MIN | 10.700 [10.700 to 10.700] | 56.200 [42.700 to 69.700]
  WEEK19 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1 | 2
  WEEK19 CROSSOVER, EOI+2HR | 4.570 [4.570 to 4.570] | 21.750 [15.400 to 28.100]
  WEEK19 CROSSOVER, EOI+4HR: number analyzed (Participants) | 0 | 2
  WEEK19 CROSSOVER, EOI+4HR |  | 9.525 [5.750 to 13.300]
  WEEK19 CROSSOVER, EOI+8HR: number analyzed (Participants) | 0 | 1
  WEEK19 CROSSOVER, EOI+8HR |  | 5.730 [5.730 to 5.730]

29. Secondary Outcome: Crossover Phase: AUC(0-tau) Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 4, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 1 | 4
h*ng/mL
  WEEK1 CROSSOVER | 3058.1703 (NA) — GCV is not estimable as only a single participant was analyzed. | 193.0653 (68.7457)
  WEEK4 CROSSOVER: number analyzed (Participants) | 0 | 3
  WEEK4 CROSSOVER |  | 201.3292 (46.6743)
  WEEK7 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER | 914.3149 (NA) — GCV is not estimable as only a single participant was analyzed. | 302.9813 (53.3033)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER | 1589.8051 (NA) — GCV is not estimable as only a single participant was analyzed. | 979.6423 (32.7400)
  WEEK13 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK13 CROSSOVER |  | 200.4303 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK19 CROSSOVER |  | 181.2630 (NA) — GCV is not estimable as only a single participant was analyzed.

30. Secondary Outcome: Crossover Phase: Cmax Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 4, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 1 | 4
ng/mL
  WEEK1 CROSSOVER | 28.900 (NA) — GCV is not estimable as only a single participant was analyzed. | 43.381 (36.411)
  WEEK4 CROSSOVER: number analyzed (Participants) | 0 | 3
  WEEK4 CROSSOVER |  | 47.379 (17.834)
  WEEK7 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER | 25.000 (NA) — GCV is not estimable as only a single participant was analyzed. | 46.371 (38.725)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER | 10.700 (NA) — GCV is not estimable as only a single participant was analyzed. | 39.435 (24.259)
  WEEK13 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK13 CROSSOVER |  | 66.300 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK19 CROSSOVER |  | 69.700 (NA) — GCV is not estimable as only a single participant was analyzed.

31. Secondary Outcome: Crossover Phase: T1/2 Following Administration of GSK3745417 in Combination With Dostarlimab (Q3W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 4, 7, 10, 13, 19
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab
Number analyzed (Participants) | 1 | 4
Hours
  WEEK1 CROSSOVER | 1016.7767 (NA) — GCV is not estimable as only a single participant was analyzed. | 15.5839 (156.6758)
  WEEK4 CROSSOVER: number analyzed (Participants) | 0 | 3
  WEEK4 CROSSOVER |  | 8.2823 (67.5066)
  WEEK7 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK7 CROSSOVER | 8.6297 (NA) — GCV is not estimable as only a single participant was analyzed. | 23.2987 (1163.1768)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1 | 2
  WEEK10 CROSSOVER | 3336.2317 (NA) — GCV is not estimable as only a single participant was analyzed. | 2.2461 (10.8792)
  WEEK13 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK13 CROSSOVER |  | 2.1918 (NA) — GCV is not estimable as only a single participant was analyzed.
  WEEK19 CROSSOVER: number analyzed (Participants) | 0 | 1
  WEEK19 CROSSOVER |  | 2.2090 (NA) — GCV is not estimable as only a single participant was analyzed.

32. Secondary Outcome: Crossover Phase: GSK3745417 Concentrations in Plasma Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Pre-dose and EOI+5min/ 2HR/4HR on crossover W 1-4, 7,10,19; EOI+15min/30 min/45 min/1HR/ 6HR/ 24HR on crossover W 1,4,7;EOI+12HR/18HR on crossover W 4;EOI+8HR on crossover W 1-4,7,10
Population: as for outcome 9
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 5
ng/mL
  WEEK1 CROSSOVER, PREDOSE | 0.000 [0.000 to 1.700]
  WEEK1 CROSSOVER, EOI+5MIN | 15.800 [10.000 to 47.100]
  WEEK1 CROSSOVER, EOI+15MIN | 14.600 [9.140 to 40.800]
  WEEK1 CROSSOVER, EOI+30MIN | 13.200 [9.210 to 24.300]
  WEEK1 CROSSOVER, EOI+45MIN | 10.700 [8.070 to 19.400]
  WEEK1 CROSSOVER, EOI+1HR | 9.530 [6.080 to 18.100]
  WEEK1 CROSSOVER, EOI+2HR | 5.780 [2.750 to 11.600]
  WEEK1 CROSSOVER, EOI+4HR | 2.520 [0.612 to 5.740]
  WEEK1 CROSSOVER, EOI+6HR | 1.130 [0.232 to 3.130]
  WEEK1 CROSSOVER, EOI+8HR | 0.507 [0.165 to 1.420]
  WEEK1 CROSSOVER, EOI+24HR | 0.000 [0.000 to 0.327]
  WEEK2 CROSSOVER, PREDOSE: number analyzed (Participants) | 3
  WEEK2 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000]
  WEEK2 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 3
  WEEK2 CROSSOVER, EOI+5MIN | 20.800 [4.390 to 23.900]
  WEEK2 CROSSOVER, EOI+2HR: number analyzed (Participants) | 4
  WEEK2 CROSSOVER, EOI+2HR | 10.040 [2.640 to 11.500]
  WEEK2 CROSSOVER, EOI+4HR: number analyzed (Participants) | 4
  WEEK2 CROSSOVER, EOI+4HR | 3.845 [1.690 to 5.340]
  WEEK2 CROSSOVER, EOI+8HR: number analyzed (Participants) | 3
  WEEK2 CROSSOVER, EOI+8HR | 0.968 [0.871 to 1.010]
  WEEK3 CROSSOVER, PREDOSE: number analyzed (Participants) | 4
  WEEK3 CROSSOVER, PREDOSE | 0.000 [0.000 to 1.020]
  WEEK3 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 3
  WEEK3 CROSSOVER, EOI+5MIN | 17.600 [14.900 to 21.200]
  WEEK3 CROSSOVER, EOI+2HR: number analyzed (Participants) | 4
  WEEK3 CROSSOVER, EOI+2HR | 9.065 [4.990 to 12.500]
  WEEK3 CROSSOVER, EOI+4HR: number analyzed (Participants) | 4
  WEEK3 CROSSOVER, EOI+4HR | 5.125 [1.850 to 7.770]
  WEEK3 CROSSOVER, EOI+8HR: number analyzed (Participants) | 3
  WEEK3 CROSSOVER, EOI+8HR | 0.826 [0.576 to 3.870]
  WEEK4 CROSSOVER, PREDOSE: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.349]
  WEEK4 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+5MIN | 15.900 [7.730 to 31.500]
  WEEK4 CROSSOVER, EOI+15MIN: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+15MIN | 14.800 [8.070 to 24.800]
  WEEK4 CROSSOVER, EOI+30MIN: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+30MIN | 12.750 [6.030 to 19.100]
  WEEK4 CROSSOVER, EOI+45MIN: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+45MIN | 11.000 [4.870 to 16.700]
  WEEK4 CROSSOVER, EOI+1HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+1HR | 10.415 [3.530 to 13.900]
  WEEK4 CROSSOVER, EOI+2HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+2HR | 6.315 [2.280 to 10.400]
  WEEK4 CROSSOVER, EOI+4HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+4HR | 2.325 [0.247 to 7.760]
  WEEK4 CROSSOVER, EOI+6HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+6HR | 0.895 [0.241 to 6.770]
  WEEK4 CROSSOVER, EOI+8HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+8HR | 0.384 [0.156 to 5.480]
  WEEK4 CROSSOVER, EOI+12HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+12HR | 0.248 [0.000 to 3.010]
  WEEK4 CROSSOVER, EOI+18HR: number analyzed (Participants) | 3
  WEEK4 CROSSOVER, EOI+18HR | 0.159 [0.000 to 1.880]
  WEEK4 CROSSOVER, EOI+24HR: number analyzed (Participants) | 4
  WEEK4 CROSSOVER, EOI+24HR | 0.055 [0.000 to 1.660]
  WEEK7 CROSSOVER, PREDOSE: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000]
  WEEK7 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+5MIN | 17.500 [11.900 to 23.100]
  WEEK7 CROSSOVER, EOI+15MIN: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+15MIN | 15.100 [10.100 to 20.100]
  WEEK7 CROSSOVER, EOI+30MIN: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+30MIN | 11.600 [7.000 to 16.200]
  WEEK7 CROSSOVER, EOI+45MIN: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+45MIN | 9.550 [5.400 to 13.700]
  WEEK7 CROSSOVER, EOI+1HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+1HR | 7.995 [4.090 to 11.900]
  WEEK7 CROSSOVER, EOI+2HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+2HR | 4.415 [1.610 to 7.220]
  WEEK7 CROSSOVER, EOI+4HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+4HR | 1.503 [0.295 to 2.710]
  WEEK7 CROSSOVER, EOI+6HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+6HR | 0.364 [0.111 to 0.616]
  WEEK7 CROSSOVER, EOI+8HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+8HR | 0.199 [0.000 to 0.398]
  WEEK7 CROSSOVER, EOI+24HR: number analyzed (Participants) | 2
  WEEK7 CROSSOVER, EOI+24HR | 0.000 [0.000 to 0.000]
  WEEK10 CROSSOVER, PREDOSE: number analyzed (Participants) | 1
  WEEK10 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000]
  WEEK10 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1
  WEEK10 CROSSOVER, EOI+5MIN | 34.700 [34.700 to 34.700]
  WEEK10 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1
  WEEK10 CROSSOVER, EOI+2HR | 13.900 [13.900 to 13.900]
  WEEK10 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1
  WEEK10 CROSSOVER, EOI+4HR | 6.430 [6.430 to 6.430]
  WEEK10 CROSSOVER, EOI+8HR: number analyzed (Participants) | 1
  WEEK10 CROSSOVER, EOI+8HR | 1.790 [1.790 to 1.790]
  WEEK19 CROSSOVER, PREDOSE: number analyzed (Participants) | 1
  WEEK19 CROSSOVER, PREDOSE | 0.000 [0.000 to 0.000]
  WEEK19 CROSSOVER, EOI+5MIN: number analyzed (Participants) | 1
  WEEK19 CROSSOVER, EOI+5MIN | 37.000 [37.000 to 37.000]
  WEEK19 CROSSOVER, EOI+2HR: number analyzed (Participants) | 1
  WEEK19 CROSSOVER, EOI+2HR | 19.300 [19.300 to 19.300]
  WEEK19 CROSSOVER, EOI+4HR: number analyzed (Participants) | 1
  WEEK19 CROSSOVER, EOI+4HR | 12.500 [12.500 to 12.500]

33. Secondary Outcome: Crossover Phase: AUC(0-tau) Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 2, 3, 4, 5, 7, 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 5
h*ng/mL
  WEEK1 CROSSOVER | 47.4854 (61.4090)
  WEEK2 CROSSOVER: number analyzed (Participants) | 4
  WEEK2 CROSSOVER | 119.0544 (129.1524)
  WEEK3 CROSSOVER: number analyzed (Participants) | 3
  WEEK3 CROSSOVER | 152.6791 (93.5753)
  WEEK4 CROSSOVER: number analyzed (Participants) | 4
  WEEK4 CROSSOVER | 45.7777 (183.4279)
  WEEK5 CROSSOVER: number analyzed (Participants) | 3
  WEEK5 CROSSOVER | 41.5618 (39.4549)
  WEEK7 CROSSOVER: number analyzed (Participants) | 2
  WEEK7 CROSSOVER | 23.9841 (110.4741)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1
  WEEK10 CROSSOVER | 81.4712 (NA) — GCV is not estimable as only a single participant was analyzed.

34. Secondary Outcome: Crossover Phase: Cmax Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 2, 3, 4, 5, 7, 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 5
ng/mL
  WEEK1 CROSSOVER | 18.932 (64.770)
  WEEK2 CROSSOVER: number analyzed (Participants) | 4
  WEEK2 CROSSOVER | 12.504 (90.216)
  WEEK3 CROSSOVER: number analyzed (Participants) | 3
  WEEK3 CROSSOVER | 13.412 (34.669)
  WEEK4 CROSSOVER: number analyzed (Participants) | 4
  WEEK4 CROSSOVER | 15.899 (60.615)
  WEEK5 CROSSOVER: number analyzed (Participants) | 3
  WEEK5 CROSSOVER | 22.354 (19.308)
  WEEK7 CROSSOVER: number analyzed (Participants) | 2
  WEEK7 CROSSOVER | 16.580 (49.604)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1
  WEEK10 CROSSOVER | 34.700 (NA) — GCV is not estimable as only a single participant was analyzed.

35. Secondary Outcome: Crossover Phase: T1/2 Following Administration of GSK3745417 in Combination With Dostarlimab (Q1W)
Description: as for outcome 16
Time Frame: Crossover Week 1, 2, 3, 4, 5, 7, 10
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
Number analyzed (Participants) | 5
Hours
  WEEK1 CROSSOVER | 2.1460 (66.2957)
  WEEK2 CROSSOVER: number analyzed (Participants) | 4
  WEEK2 CROSSOVER | 4.7086 (327.1693)
  WEEK3 CROSSOVER: number analyzed (Participants) | 3
  WEEK3 CROSSOVER | 2.1828 (54.2570)
  WEEK4 CROSSOVER: number analyzed (Participants) | 4
  WEEK4 CROSSOVER | 3.7809 (121.5012)
  WEEK5 CROSSOVER: number analyzed (Participants) | 3
  WEEK5 CROSSOVER | 1.4489 (22.9248)
  WEEK7 CROSSOVER: number analyzed (Participants) | 2
  WEEK7 CROSSOVER | 1.1078 (38.4294)
  WEEK10 CROSSOVER: number analyzed (Participants) | 1
  WEEK10 CROSSOVER | 1.9742 (NA) — GCV is not estimable as only a single participant was analyzed.

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to approximately 62 weeks for part 1A, up to approximately 93 weeks for part 2A and up to 30.3 weeks for crossover phase.
Description: All treated population included all the participants who received at least one dose of GSK3745417.
Arm/Group | Part 1A: GSK3745417 0.1 mg (Q3W) | Part 1A: GSK3745417 0.2 mg (Q3W) | Part 1A: GSK3745417 0.1 mg (Q1W) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) | Part 1A: GSK3745417 0.2 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab
All-Cause Mortality (participants affected / at risk) | 3/3 | 5/6 | 6/14 | 0/2 | 14/19 | 7/10 | 8/9 | 3/4 | 8/12 | 4/4 | 2/3 | 8/10 | 0/1 | 0/1 | 1/4 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 4/14 | 0/2 | 7/19 | 3/10 | 2/9 | 1/4 | 6/12 | 3/4 | 2/3 | 4/10 | 1/1 | 0/1 | 1/4 | 1/5
Other Adverse Events (participants affected / at risk) | 2/3 | 5/6 | 14/14 | 2/2 | 19/19 | 10/10 | 9/9 | 4/4 | 12/12 | 4/4 | 3/3 | 10/10 | 1/1 | 1/1 | 3/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: GSK3745417 0.1 mg (Q3W) (N=3) | Part 1A: GSK3745417 0.2 mg (Q3W) (N=6) | Part 1A: GSK3745417 0.1 mg (Q1W) (N=14) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) (N=2) | Part 1A: GSK3745417 0.2 mg (Q1W) (N=19) | Part 1A: GSK3745417 0.4 mg (Q1W) (N=10) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis (N=9) | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab (N=4) | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab (N=12) | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=4) | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=3) | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab (N=10) | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab (N=1) | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab (N=1) | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab (N=4) | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A: GSK3745417 0.1 mg (Q3W) (N=3) | Part 1A: GSK3745417 0.2 mg (Q3W) (N=6) | Part 1A: GSK3745417 0.1 mg (Q1W) (N=14) | Part 1A: Japan GSK3745417 0.1 mg (Q1W) (N=2) | Part 1A: GSK3745417 0.2 mg (Q1W) (N=19) | Part 1A: GSK3745417 0.4 mg (Q1W) (N=10) | Part 1A: GSK3745417 0.4 mg (Q1W) Prophylaxis (N=9) | Part 2A: GSK3745417 0.1 mg (Q3W) + Dostarlimab (N=4) | Part 2A: GSK3745417 0.2 mg (Q3W) + Dostarlimab (N=12) | Part 2A: GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=4) | Part 2A: Imaging GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=3) | Part 2A: GSK3745417 0.2 mg (Q1W) + Dostarlimab (N=10) | Part 2A: Imaging GSK3745417 0.2 mg (Q1W) + Dostarlimab (N=1) | Crossover: GSK3745417 0.1 mg (Q3W) + Dostarlimab (N=1) | Crossover: GSK3745417 0.2 mg (Q3W) + Dostarlimab (N=4) | Crossover: GSK3745417 0.1 mg (Q1W) + Dostarlimab (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 7 (10) | 0 (0) | 4 (10) | 3 (10) | 5 (8) | 0 (0) | 2 (3) | 0 (0) | 2 (7) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 1 (2)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 4 (17) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 3 (13) | 7 (17) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (11) | 5 (6) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 3 (5) | 4 (6) | 0 (0) | 7 (24) | 10 (69) | 6 (19) | 0 (0) | 4 (7) | 2 (2) | 2 (2) | 5 (14) | 1 (3) | 0 (0) | 2 (5) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 6 (7) | 0 (0) | 10 (21) | 5 (15) | 7 (12) | 1 (2) | 6 (6) | 2 (4) | 1 (1) | 4 (6) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (8) | 4 (11) | 1 (1) | 13 (39) | 10 (56) | 6 (26) | 0 (0) | 8 (13) | 3 (3) | 2 (4) | 7 (8) | 1 (3) | 1 (5) | 2 (7) | 1 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (14) | 5 (11) | 4 (7) | 0 (0) | 4 (7) | 1 (1) | 1 (1) | 5 (6) | 1 (2) | 0 (0) | 1 (5) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (5) | 3 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 3 (5) | 0 (0) | 7 (12) | 5 (24) | 1 (2) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 1 (1) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (8) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurodesis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (8) | 3 (5) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT03843359/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03843359/SAP_001.pdf